CLINICAL TRIAL: NCT02108171
Title: A Randomised Controlled Trial of Intranasal Dexmedetomidine as Premedication for Suspension Laryngoscopy
Brief Title: Intranasal Dexmedetomidine Premedication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, Xiangcai Ruan, MD, PhD, Vice-Director in Dept Anesth & Pain, Vice Chair, Guangzhou First People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GZFPH-IRB-2013-086
Record Dates: First submitted 2014-03-30; First posted 2014-04-09 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Benign Neoplasm of Vocal Fold - Glottis
Keywords: intranasal; dexmedetomidine; early recovery; suspension laryngoscopy
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dexmedetomidine (Active Comparator): intranasal dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- placebo (Placebo Comparator): intranasal saline
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dexmedetomidine — intranasal dexmedetomidine 1μg.kg-1，0.9% saline was added to make a final volume of 1 mL.all patients received intranasal medication at approximately 45-60 min before induction of anesthesia.
  Other Names: intranasal dexmedetomidine
  Arms: dexmedetomidine
Drug: placebo — 0.9% saline 1 mL all patients received intranasal medication at approximately 45-60 min before induction of anesthesia.
  Other Names: saline
  Arms: placebo

SUMMARY:
Most patients with preoperative varying degrees of stress, anxiety, which makes the stress response in patients and affect the normal conduct of anesthesia and surgery.The sympathetic system hyperexcitability prone to cause adverse cardiovascular events and affect postoperative recovery. However, phenobarbital, as the traditional premedication, has less sedative, weak anxiolytic and other shortcomings. Midazolam accompanied by inhibition of respiration,excessive sedation, easily induced delirium,prolonged recovery time and so on. Dexmedetomidine is a highly selective α2-adrenergic receptor agonist, it has sedative, anxiolytic, no inhibition of respiration, and also colorless, odorless, non-mucosal stimulation, nasal drip ease of administration, patient acceptance, comfortable. Therefore, dexmedetomidine as premedication has certain advantages. The purpose of this research is to study sedative effect, safety and the impact of anesthesia recovery period of intranasal dexmedetomidine premedication for suspension laryngoscopy.

DETAILED DESCRIPTION:
All patients received intranasal dexmedetomidine (1μg.kg-1) or placebo at approximately 45 min before induction of anesthesia.The study drug was prepared in a 1-ml syringe.An equal volume of dexmedetomidine or placebo was dropped into each nostril by a blinded research assistant in the supine position.Automatic sphygmomanometer measure blood pressure.Oxygen saturation and heart rate were measured by a pulse oximeter. Respiratory rate, sedation score and anxiety levels regularly assessed. Patients with general anesthesia, suspension laryngoscopy surgery and postoperative care, standard monitoring are unified.

ELIGIBILITY:
Inclusion Criteria:

* Surgery:The laryngoscope vocal polyp excision
* Aged 18 to 60 years old
* Body mass index (BMI) < 30 kg/m2
* American society of Anesthesiologist (ASA) I -II

Exclusion Criteria:

* The investigator refused to participate
* Known allergy or hypersensitive reaction to dexmedetomidine or anesthetic
* With previous history of heart disease
* Pregnant women; no reliable contraceptive measures in postmenopausal women
* Preoperative heart rate less than 45bpm; Ⅱ or Ⅲ degree atrioventricular block; ischemic heart disease
* Taking antihypertensive drugs such as methyldopa, clonidine and other α2 receptor agonist
* Asthma
* Sleep apnea syndrome
* Liver and kidney dysfunction
* Known to suffer from mental illness
* Long-term use of sedatives and analgesics in patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiangcai Ruan, MD, PHD, Principal Investigator — Guangzhou First Municipal People's Hospital,Guangzhou Medical College
Locations (2):
- China (2):
  - Guangzhou First Municipal People's Hospital, Guangzhou, Guangdong
  - Guangzhou First Municipal People's Hospital, Guangzhou

REFERENCES:
- [Background] Sheta SA, Al-Sarheed MA, Abdelhalim AA. Intranasal dexmedetomidine vs midazolam for premedication in children undergoing complete dental rehabilitation: a double-blinded randomized controlled trial. Paediatr Anaesth. 2014 Feb;24(2):181-9. doi: 10.1111/pan.12287. Epub 2013 Nov 15. PMID 24237879
- [Background] Yuen VM, Irwin MG, Hui TW, Yuen MK, Lee LH. A double-blind, crossover assessment of the sedative and analgesic effects of intranasal dexmedetomidine. Anesth Analg. 2007 Aug;105(2):374-80. doi: 10.1213/01.ane.0000269488.06546.7c. PMID 17646493
- [Background] Yuen VM, Hui TW, Irwin MG, Yao TJ, Chan L, Wong GL, Shahnaz Hasan M, Shariffuddin II. A randomised comparison of two intranasal dexmedetomidine doses for premedication in children. Anaesthesia. 2012 Nov;67(11):1210-6. doi: 10.1111/j.1365-2044.2012.07309.x. Epub 2012 Sep 5. PMID 22950484
- [Background] Cheung CW, Ng KF, Liu J, Yuen MY, Ho MH, Irwin MG. Analgesic and sedative effects of intranasal dexmedetomidine in third molar surgery under local anaesthesia. Br J Anaesth. 2011 Sep;107(3):430-7. doi: 10.1093/bja/aer164. Epub 2011 Jun 16. PMID 21685111
- [Background] Iirola T, Vilo S, Manner T, Aantaa R, Lahtinen M, Scheinin M, Olkkola KT. Bioavailability of dexmedetomidine after intranasal administration. Eur J Clin Pharmacol. 2011 Aug;67(8):825-31. doi: 10.1007/s00228-011-1002-y. Epub 2011 Feb 12. PMID 21318594
- [Background] Nooh N, Sheta SA, Abdullah WA, Abdelhalim AA. Intranasal atomized dexmedetomidine for sedation during third molar extraction. Int J Oral Maxillofac Surg. 2013 Jul;42(7):857-62. doi: 10.1016/j.ijom.2013.02.003. Epub 2013 Mar 14. PMID 23497981
- [Background] Ambi US, Joshi C, Ganeshnavar A, Adarsh E. Intranasal dexmedetomidine for paediatric sedation for diagnostic magnetic resonance imaging studies. Indian J Anaesth. 2012 Nov;56(6):587-8. doi: 10.4103/0019-5049.104588. No abstract available. PMID 23325950
- [Background] Yuen VM, Hui TW, Irwin MG, Yao TJ, Wong GL, Yuen MK. Optimal timing for the administration of intranasal dexmedetomidine for premedication in children. Anaesthesia. 2010 Sep;65(9):922-9. doi: 10.1111/j.1365-2044.2010.06453.x. PMID 20645951
- [Derived] Lu C, Zhang LM, Zhang Y, Ying Y, Li L, Xu L, Ruan X. Intranasal Dexmedetomidine as a Sedative Premedication for Patients Undergoing Suspension Laryngoscopy: A Randomized Double-Blind Study. PLoS One. 2016 May 19;11(5):e0154192. doi: 10.1371/journal.pone.0154192. eCollection 2016. PMID 27196121

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients of ASA physical status I or II, aged between 18 and 60 yrs, scheduled for elective suspension for remove of benign lesions under general anesthesia between September 2013 and April 2014
Pre-assignment Details: 40 patients receive intranasal dexmedetomidine (1 µg.kg-1 in 1 ml) and 41 patients receive intranasal saline (1 ml) 45-60 min before anesthetic induction.
Period: Overall Study
Arm/Group | Dexmedetomidine | Placebo
Started | 40 | 41
Completed | 40 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Placebo | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 41 | 81
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (10.1) | 43.6 (9.2) | 44.75 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 28 | 52
  Male | 16 | 13 | 29
BMI [Mean (Standard Deviation); unit: kg per square meter] | 22.49 (3.03) | 22.75 (3.07) | 22.62 (3.04)
Weight [Mean (Standard Deviation); unit: kg] | 59.4 (9.1) | 60.1 (10.4) | 59.76 (9.7)
Height [Mean (Standard Deviation); unit: cm] | 162.5 (8.0) | 162.2 (6.1) | 162.4 (7.1)
Duration time [Mean (Standard Deviation); unit: min]
  from drug administration to arrival at OR | 42.3 (20.4) | 39.3 (18.2) | 40.8 (19.2)
  from drug administration to intubation | 62.1 (23.4) | 60.8 (18.9) | 61.5 (21.2)
  Duration of surgery | 21.4 (14.1) | 26.1 (24.7) | 23.7 (20.1)

OUTCOME MEASURES:

1. Primary Outcome: Extubation Time After Intranasal Dexmedetomidine Premedication
Description: The times from stopping anesthetic infusions to adequate ventilation, consciousness and extubation after intranasal dexmedetomidine or placebo administration
Time Frame: 1 days
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 40 | 41
min
  Extubation time | 18.58 (7.376) | 17.16 (7.142)
  consciousness time | 16.21 (6.278) | 14.74 (6.353)
  adequate ventilation time | 8.24 (3.183) | 7.87 (2.648)

2. Secondary Outcome: Modified OAA/S Scores of Patients Receiving Intranasal Placebo or Dexmedetomidine
Description: Modified Observer's Assessment of Alertness/Sedation scale (OAA/S) scores and 4 point anxiety score of patients receiving intranasal placebo or dexmedetomidine.
  Modified Observer's Assessment of Alertness/Sedation Scale:
  6 Appears alert and awake, responds readily to name spoken in normal tone 5 Appears asleep but responds readily to name spoken in normal tone 4 Lethargic response to name spoken in normal tone 3 Responds only after name is called loudly or repeatedly 2 Responds only after mild prodding or shaking
  1 Does not respond to mild prodding or shaking 0 Does not respond to noxious stimulus.
Time Frame: 1 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 40 | 41
units on a scale
  Before intranasal drugs | 6 [6 to 6] | 6 [6 to 6]
  Pre-induction | 4 [4 to 5] | 6 [5 to 6]
  After extubation | 4 [3 to 4] | 4 [3 to 5]

3. Secondary Outcome: Heart Rate (HR) of Patients Receiving Intranasal Placebo or Dexmedetomidine
Description: Heart rate (HR) of patients receiving intranasal placebo or dexmedetomidine. HR was monitored in the study.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 40 | 41
bpm
  Before intranasal drops | 71.75 (1.493) | 72.2 (2.105)
  On arrival at operating room | 66.93 (1.732) | 71.53 (1.780)
  At pre-induction | 65.63 (1.502) | 72 (1.721)
  After tracheal intubation | 70.62 (12.13) | 85.26 (16.93)
  After inserting operative laryngoscope | 75.48 (16.55) | 83.61 (18.34)
  After removal of laryngoscope | 71.76 (9.73) | 77.06 (11.52)
  On arrival at PACU | 67.14 (9.08) | 68.9 (10.94)
  At emergency | 67.81 (11.85) | 72.48 (13.45)
  After tracheal extubation | 64.24 (13.19) | 73.65 (15.5)
  Before leaving PACU | 65.52 (9.21) | 69.32 (10.04)

4. Other Pre Specified Outcome: Baseline Characteristic Data (Weight) of Patients Receiving Intranasal Placebo
Description: Baseline characteristic data of patients receiving intranasal placebo The weights of 41 adult patients receiving intranasal placebo
Time Frame: 1 day
Measure: Number; unit: kg
Arm/Group | Placebo
Number analyzed (Participants) | 41
kg
  Patient number1 | 54
  Patient number4 | 67
  Patient number8 | 80
  Patient number12 | 80
  Patient number13 | 65
  Patient number14 | 49
  Patient number15 | 60
  Patient number16 | 55
  Patient number17 | 73
  Patient number19 | 59
  Patient number20 | 71.5
  Patient number21 | 59
  Patient number22 | 57
  Patient number23 | 55
  Patient number26 | 59
  Patient number27 | 53
  Patient number30 | 45
  Patient number32 | 53
  Patient number34 | 58
  Patient number35 | 78
  Patient number37 | 65
  Patient number39 | 69
  Patient number41 | 47
  Patient number42 | 61
  Patient number43 | 50
  Patient number45 | 40
  Patient number47 | 55
  Patient number48 | 51
  Patient number49 | 50
  Patient number51 | 71
  Patient number54 | 69
  Patient number55 | 79
  Patient number60 | 60
  Patient number64 | 54
  Patient number68 | 47
  Patient number69 | 51
  Patient number70 | 60
  Patient number73 | 60
  Patient number77 | 57
  Patient number78 | 61
  Patient number81 | 78

5. Other Pre Specified Outcome: Baseline Characteristic Data (Weight) of Patients Receiving Intranasal Dexmedetomidine
Description: Baseline characteristic data of patients receiving intranasal dexmedetomidine The weights of 40 adult patients receiving intranasal dexmedetomidine
Time Frame: 1 day
Measure: Number; unit: kg
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
kg
  Patient number2 | 61
  Patient number3 | 50
  Patient number5 | 58
  Patient number6 | 52
  Patient number7 | 64
  Patient number9 | 62
  Patient number10 | 56
  Patient number11 | 53
  Patient number18 | 59
  Patient number24 | 54
  Patient number25 | 65
  Patient number28 | 68
  Patient number29 | 58
  Patient number31 | 78
  Patient number33 | 53
  Patient number36 | 75
  Patient number38 | 75
  Patient number40 | 59
  Patient number44 | 73
  Patient number46 | 56
  Patient number50 | 46
  Patient number52 | 54
  Patient number53 | 47.5
  Patient number56 | 75
  Patient number57 | 80
  Patient number58 | 69
  Patient number59 | 57
  Patient number61 | 65
  Patient number62 | 58
  Patient number63 | 60
  Patient number65 | 45
  Patient number66 | 52
  Patient number67 | 45
  Patient number71 | 52
  Patient number72 | 52
  Patient number74 | 58
  Patient number75 | 60
  Patient number76 | 50
  Patient number79 | 60
  Patient number80 | 72

6. Other Pre Specified Outcome: Baseline Characteristic Data (Height) of Patients Receiving Intranasal Placebo
Description: Baseline characteristic data of patients receiving intranasal placebo The heights of 41 adult patients receiving intranasal placebo
Time Frame: 1 day
Measure: Number; unit: cm
Arm/Group | Placebo
Number analyzed (Participants) | 41
cm
  Patient number1 | 163
  Patient number4 | 171
  Patient number8 | 177
  Patient number12 | 170
  Patient number13 | 168
  Patient number14 | 155
  Patient number15 | 160
  Patient number16 | 165
  Patient number17 | 165
  Patient number19 | 163
  Patient number20 | 162
  Patient number21 | 157
  Patient number22 | 160
  Patient number23 | 159
  Patient number26 | 157
  Patient number27 | 168
  Patient number30 | 168
  Patient number32 | 160
  Patient number34 | 162
  Patient number35 | 165
  Patient number37 | 170
  Patient number39 | 161
  Patient number41 | 160
  Patient number42 | 154
  Patient number43 | 157
  Patient number45 | 150
  Patient number47 | 156
  Patient number48 | 155
  Patient number49 | 160
  Patient number51 | 173
  Patient number54 | 169
  Patient number55 | 165
  Patient number60 | 162
  Patient number64 | 155
  Patient number68 | 155
  Patient number69 | 164
  Patient number70 | 163
  Patient number73 | 162
  Patient number77 | 160
  Patient number78 | 154
  Patient number81 | 172

7. Other Pre Specified Outcome: Baseline Characteristic Data (Height) of Patients Receiving Intranasal Dexmedetomidine
Description: Baseline characteristic data of patients receiving intranasal dexmedetomidine The heights of 40 adult patients receiving intranasal placebo
Time Frame: 1 day
Measure: Number; unit: cm
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
cm
  Patient number2 | 163
  Patient number3 | 155
  Patient number5 | 182
  Patient number6 | 169
  Patient number7 | 160
  Patient number9 | 150
  Patient number10 | 170
  Patient number11 | 158
  Patient number18 | 160
  Patient number24 | 165
  Patient number25 | 167
  Patient number28 | 170
  Patient number29 | 160
  Patient number31 | 167
  Patient number33 | 150
  Patient number36 | 162
  Patient number38 | 170
  Patient number40 | 160
  Patient number44 | 157
  Patient number46 | 160
  Patient number50 | 150
  Patient number52 | 151
  Patient number53 | 160
  Patient number56 | 176
  Patient number57 | 165
  Patient number58 | 172
  Patient number59 | 152
  Patient number61 | 174
  Patient number62 | 156
  Patient number63 | 167
  Patient number65 | 154
  Patient number66 | 155
  Patient number67 | 156
  Patient number71 | 157
  Patient number72 | 157
  Patient number74 | 167
  Patient number75 | 167
  Patient number76 | 161
  Patient number79 | 174
  Patient number80 | 173

8. Other Pre Specified Outcome: Baseline Characteristics (Sex)of Patients Receiving Intranasal Placebo or Dexmedetomidine
Description: Baseline characteristics (sex)of patients receiving intranasal placebo or dexmedetomidine The sex of 81 adult patients receiving intranasal placebo or dexmedetomidine
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 40 | 41
participants
  Male | 16 | 13
  Female | 24 | 28

9. Other Pre Specified Outcome: Baseline Characteristics (ASA Status) of Patients Receiving Intranasal Placebo or Dexmedetomidine
Description: American Society of Anesthesiologists (ASA) status of patients receiving intranasal placebo or dexmedetomidine.
  ASA I: No organic, physiologic, biochemical or psychiatric disturbance ASA II: A patient with mild systemic disease that results in no functional limitation.
  ASA III: A patient with severe systemic disease that results in functional impairment.
  ASA IV: Severe systemic disease that is a constant threat to life. ASA V: Moribund condition in a patient who is not expected to survive with or without the operation.
  ASA VI: Declared brain death patient whose organs are being harvested for transplantation.
Time Frame: 1 day
Measure: Number; unit: participant
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 40 | 41
participant
  ASA I | 36 | 38
  ASA II | 4 | 3
  ASA III | 0 | 0
  ASA IV | 0 | 0
  ASA V | 0 | 0
  ASA VI | 0 | 0

10. Other Pre Specified Outcome: Duration From Intranasal Drug Administration to Arrival at Operating Room of Patients Receiving Intranasal Placebo
Description: Duration from intranasal drug administration to arrival at operating room of patients receiving intranasal placebo surgical data of patients receiving intranasal placebo
Time Frame: 1 day
Measure: Number; unit: minutes
Arm/Group | Placebo
Number analyzed (Participants) | 41
minutes
  Patient number1 | 50
  Patient number4 | 45
  Patient number8 | 60
  Patient number12 | 30
  Patient number13 | 45
  Patient number14 | 45
  Patient number15 | 65
  Patient number16 | 75
  Patient number17 | 78
  Patient number19 | 35
  Patient number20 | 60
  Patient number21 | 60
  Patient number22 | 40
  Patient number23 | 0
  Patient number26 | 33
  Patient number27 | 35
  Patient number30 | 0
  Patient number32 | 40
  Patient number34 | 35
  Patient number35 | 45
  Patient number37 | 40
  Patient number39 | 55
  Patient number41 | 40
  Patient number42 | 40
  Patient number43 | 18
  Patient number45 | 15
  Patient number47 | 30
  Patient number48 | 35
  Patient number49 | 0
  Patient number51 | 40
  Patient number54 | 5
  Patient number55 | 40
  Patient number60 | 45
  Patient number64 | 27
  Patient number68 | 50
  Patient number69 | 40
  Patient number70 | 52
  Patient number73 | 45
  Patient number77 | 40
  Patient number78 | 40
  Patient number81 | 40

11. Other Pre Specified Outcome: Duration From Intranasal Drug Administration to Arrival at Operating Room of Patients Receiving Intranasal Dexmedetomidine
Description: Duration From Intranasal Drug Administration to Arrival at Operating Room of Patients Receiving Intranasal dexmedetomidine surgical data of patients receiving intranasal dexmedetomidine
Time Frame: 1 day
Measure: Number; unit: minutes
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
minutes
  Patient number2 | 100
  Patient number3 | 35
  Patient number5 | 40
  Patient number6 | 45
  Patient number7 | 40
  Patient number9 | 41
  Patient number10 | 35
  Patient number11 | 35
  Patient number18 | 95
  Patient number24 | 40
  Patient number25 | 40
  Patient number28 | 30
  Patient number29 | 40
  Patient number31 | 30
  Patient number33 | 5
  Patient number36 | 5
  Patient number38 | 6
  Patient number40 | 75
  Patient number44 | 40
  Patient number46 | 32
  Patient number50 | 5
  Patient number52 | 45
  Patient number53 | 65
  Patient number56 | 38
  Patient number57 | 38
  Patient number58 | 30
  Patient number59 | 25
  Patient number61 | 60
  Patient number62 | 50
  Patient number63 | 62
  Patient number65 | 44
  Patient number66 | 47
  Patient number67 | 55
  Patient number71 | 60
  Patient number72 | 50
  Patient number74 | 60
  Patient number75 | 45
  Patient number76 | 43
  Patient number79 | 32
  Patient number80 | 30

12. Other Pre Specified Outcome: Duration From Intranasal Drug Administration to Anesthesia Intubation of Patients Receiving Intranasal Placebo
Description: Duration from intranasal drug administration to anesthesia intubation of Patients Receiving Intranasal Placebo surgical data of patients receiving intranasal placebo
Time Frame: 1 day
Measure: Number; unit: minutes
Arm/Group | Placebo
Number analyzed (Participants) | 41
minutes
  Patient number1 | 60
  Patient number4 | 77
  Patient number8 | 96
  Patient number12 | 48
  Patient number13 | 54
  Patient number14 | 55
  Patient number15 | 77
  Patient number16 | 83
  Patient number17 | 84
  Patient number19 | 54
  Patient number20 | 70
  Patient number21 | 73
  Patient number22 | 45
  Patient number23 | 48
  Patient number26 | 45
  Patient number27 | 45
  Patient number30 | 50
  Patient number32 | 48
  Patient number34 | 51
  Patient number35 | 47
  Patient number37 | 47
  Patient number39 | 69
  Patient number41 | 54
  Patient number42 | 49
  Patient number43 | 46
  Patient number45 | 23
  Patient number47 | 40
  Patient number48 | 79
  Patient number49 | 57
  Patient number51 | 49
  Patient number54 | 53
  Patient number55 | 54
  Patient number60 | 69
  Patient number64 | 115
  Patient number68 | 62
  Patient number69 | 113
  Patient number70 | 68
  Patient number73 | 71
  Patient number77 | 54
  Patient number78 | 51
  Patient number81 | 54

13. Other Pre Specified Outcome: Duration From Intranasal Drug Administration to Anesthesia Intubation of Patients Receiving Intranasal Dexmedetomidine
Description: Duration of minutes From Intranasal Drug Administration to Anesthesia Intubation of Patients Receiving Intranasal dexmedetomidine surgical data of Patients Receiving Intranasal dexmedetomidine.
Time Frame: 1 day
Measure: Number; unit: minutes
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
minutes
  Patient number2 | 112
  Patient number3 | 40
  Patient number5 | 52
  Patient number6 | 56
  Patient number7 | 50
  Patient number9 | 49
  Patient number10 | 45
  Patient number11 | 45
  Patient number18 | 105
  Patient number24 | 53
  Patient number25 | 47
  Patient number28 | 105
  Patient number29 | 45
  Patient number31 | 32
  Patient number33 | 55
  Patient number36 | 52
  Patient number38 | 46
  Patient number40 | 81
  Patient number44 | 46
  Patient number46 | 41
  Patient number50 | 52
  Patient number52 | 55
  Patient number53 | 101
  Patient number56 | 54
  Patient number57 | 45
  Patient number58 | 43
  Patient number59 | 33
  Patient number61 | 78
  Patient number62 | 60
  Patient number63 | 88
  Patient number65 | 63
  Patient number66 | 62
  Patient number67 | 69
  Patient number71 | 141
  Patient number72 | 74
  Patient number74 | 73
  Patient number75 | 61
  Patient number76 | 62
  Patient number79 | 55
  Patient number80 | 58

14. Other Pre Specified Outcome: Duration of Anesthesia of Patients Receiving Intranasal Placebo
Description: Duration of anesthesia of patients receiving intranasal placebo Duration from anesthesia intubation to anesthesia ending
Time Frame: 1 day
Measure: Number; unit: minutes
Arm/Group | Placebo
Number analyzed (Participants) | 41
minutes
  Patient number1 | 45
  Patient number4 | 33
  Patient number8 | 26
  Patient number12 | 37
  Patient number13 | 45
  Patient number14 | 34
  Patient number15 | 18
  Patient number16 | 37
  Patient number17 | 54
  Patient number19 | 48
  Patient number20 | 40
  Patient number21 | 29
  Patient number22 | 31
  Patient number23 | 32
  Patient number26 | 158
  Patient number27 | 38
  Patient number30 | 41
  Patient number32 | 30
  Patient number34 | 28
  Patient number35 | 28
  Patient number37 | 43
  Patient number39 | 35
  Patient number41 | 40
  Patient number42 | 28
  Patient number43 | 34
  Patient number45 | 69
  Patient number47 | 40
  Patient number48 | 56
  Patient number49 | 43
  Patient number51 | 78
  Patient number54 | 54
  Patient number55 | 38
  Patient number60 | 88
  Patient number64 | 38
  Patient number68 | 31
  Patient number69 | 106
  Patient number70 | 29
  Patient number73 | 31
  Patient number77 | 21
  Patient number78 | 49
  Patient number81 | 60

15. Other Pre Specified Outcome: Duration of Anesthesia of Patients Receiving Intranasal Dexmedetomidine
Description: Duration of anesthesia of patients receiving intranasal dexmedetomidine Duration from anesthesia intubation to anesthesia ending
Time Frame: 1 day
Measure: Number; unit: minutes
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
minutes
  Patient number2 | 42
  Patient number3 | 28
  Patient number5 | 87
  Patient number6 | 53
  Patient number7 | 16
  Patient number9 | 73
  Patient number10 | 36
  Patient number11 | 30
  Patient number18 | 27
  Patient number24 | 24
  Patient number25 | 49
  Patient number28 | 35
  Patient number29 | 29
  Patient number31 | 37
  Patient number33 | 27
  Patient number36 | 31
  Patient number38 | 34
  Patient number40 | 36
  Patient number44 | 48
  Patient number46 | 31
  Patient number50 | 53
  Patient number52 | 37
  Patient number53 | 29
  Patient number56 | 31
  Patient number57 | 35
  Patient number58 | 80
  Patient number59 | 49
  Patient number61 | 52
  Patient number62 | 45
  Patient number63 | 30
  Patient number65 | 28
  Patient number66 | 17
  Patient number67 | 36
  Patient number71 | 50
  Patient number72 | 24
  Patient number74 | 31
  Patient number75 | 26
  Patient number76 | 25
  Patient number79 | 44
  Patient number80 | 72

16. Other Pre Specified Outcome: Duration of Surgery of Patients Receiving Intranasal Placebo
Description: Duration of surgery of patients receiving intranasal placebo Duration from surgery beginning to anesthesia ending
Time Frame: 1 day
Measure: Number; unit: minutes
Arm/Group | Placebo
Number analyzed (Participants) | 41
minutes
  Patient number1 | 30
  Patient number4 | 19
  Patient number8 | 10
  Patient number12 | 13
  Patient number13 | 29
  Patient number14 | 14
  Patient number15 | 5
  Patient number16 | 18
  Patient number17 | 20
  Patient number19 | 56
  Patient number20 | 19
  Patient number21 | 12
  Patient number22 | 11
  Patient number23 | 10
  Patient number26 | 132
  Patient number27 | 18
  Patient number30 | 16
  Patient number32 | 11
  Patient number34 | 9
  Patient number35 | 16
  Patient number37 | 25
  Patient number39 | 12
  Patient number41 | 18
  Patient number42 | 9
  Patient number43 | 13
  Patient number45 | 48
  Patient number47 | 21
  Patient number48 | 30
  Patient number49 | 25
  Patient number51 | 60
  Patient number54 | 29
  Patient number55 | 18
  Patient number60 | 58
  Patient number64 | 19
  Patient number68 | 17
  Patient number69 | 90
  Patient number70 | 10
  Patient number73 | 16
  Patient number77 | 8
  Patient number78 | 31
  Patient number81 | 28

17. Other Pre Specified Outcome: Duration of Surgery of Patients Receiving Intranasal Dexmedetomidine
Description: Duration of surgery of patients receiving intranasal dexmedetomidine. Duration from surgery beginning to anesthesia ending
Time Frame: 1 day
Measure: Number; unit: minutes
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
minutes
  Patient number2 | 19
  Patient number3 | 14
  Patient number5 | 61
  Patient number6 | 34
  Patient number7 | 4
  Patient number9 | 50
  Patient number10 | 22
  Patient number11 | 15
  Patient number18 | 13
  Patient number24 | 10
  Patient number25 | 27
  Patient number28 | 13
  Patient number29 | 9
  Patient number31 | 19
  Patient number33 | 9
  Patient number36 | 7
  Patient number38 | 18
  Patient number40 | 20
  Patient number44 | 34
  Patient number46 | 10
  Patient number50 | 30
  Patient number52 | 24
  Patient number53 | 16
  Patient number56 | 16
  Patient number58 | 61
  Patient number57 | 18
  Patient number59 | 29
  Patient number61 | 27
  Patient number62 | 25
  Patient number63 | 11
  Patient number65 | 12
  Patient number66 | 7
  Patient number67 | 21
  Patient number71 | 33
  Patient number72 | 9
  Patient number74 | 15
  Patient number75 | 9
  Patient number76 | 7
  Patient number79 | 29
  Patient number80 | 45

18. Other Pre Specified Outcome: Modified OAA/S Score of Patients Receiving Intranasal Placebo Before Intranasal Drugs
Description: Modified OAA/S score of patients receiving intranasal placebo Before intranasal drugs Modified Observer's Assessment of Alertness/Sedation Scale (Modified OAA/S score) 6 Appears alert and awake, responds readily to name spoken in normal tone 5 Appears asleep but responds readily to name spoken in normal tone 4 Lethargic response to name spoken in normal tone 3 Responds only after name is called loudly or repeatedly 2 Responds only after mild prodding or shaking
  1 Does not respond to mild prodding or shaking 0 Does not respond to noxious stimulus
Time Frame: 1 day
Measure: Number; unit: units on a scale
Arm/Group | Placebo
Number analyzed (Participants) | 41
units on a scale
  Patient number1 | 6
  Patient number4 | 6
  Patient number8 | 6
  Patient number12 | 6
  Patient number13 | 6
  Patient number14 | 6
  Patient number15 | 6
  Patient number16 | 6
  Patient number17 | 6
  Patient number19 | 6
  Patient number20 | 6
  Patient number21 | 6
  Patient number22 | 6
  Patient number23 | 6
  Patient number26 | 6
  Patient number27 | 6
  Patient number30 | 6
  Patient number32 | 6
  Patient number34 | 6
  Patient number35 | 6
  Patient number37 | 6
  Patient number39 | 6
  Patient number41 | 6
  Patient number42 | 6
  Patient number43 | 6
  Patient number45 | 6
  Patient number47 | 6
  Patient number48 | 6
  Patient number49 | 6
  Patient number51 | 6
  Patient number54 | 6
  Patient number55 | 6
  Patient number60 | 6
  Patient number64 | 6
  Patient number68 | 6
  Patient number69 | 6
  Patient number70 | 6
  Patient number73 | 6
  Patient number77 | 6
  Patient number81 | 6
  Patient number78 | 6

19. Other Pre Specified Outcome: Modified OAA/S Score of Patients Receiving Intranasal Dexmedetomidine Before Intranasal Drugs
Description: Modified OAA/S score of patients receiving intranasal dexmedetomidine Before intranasal drugs Modified Observer's Assessment of Alertness/Sedation Scale (Modified OAA/S score) 6 Appears alert and awake, responds readily to name spoken in normal tone 5 Appears asleep but responds readily to name spoken in normal tone 4 Lethargic response to name spoken in normal tone 3 Responds only after name is called loudly or repeatedly 2 Responds only after mild prodding or shaking
  1 Does not respond to mild prodding or shaking 0 Does not respond to noxious stimulus
Time Frame: 1 day
Measure: Number; unit: units on a scale
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
units on a scale
  Patient number2 | 6
  Patient number3 | 6
  Patient number5 | 6
  Patient number6 | 6
  Patient number7 | 6
  Patient number9 | 6
  Patient number10 | 6
  Patient number11 | 6
  Patient number18 | 6
  Patient number24 | 6
  Patient number25 | 6
  Patient number28 | 6
  Patient number29 | 6
  Patient number31 | 6
  Patient number33 | 6
  Patient number36 | 6
  Patient number38 | 6
  Patient number40 | 6
  Patient number44 | 6
  Patient number46 | 6
  Patient number50 | 6
  Patient number52 | 6
  Patient number53 | 6
  Patient number56 | 6
  Patient number57 | 6
  Patient number58 | 6
  Patient number59 | 6
  Patient number61 | 6
  Patient number62 | 6
  Patient number63 | 6
  Patient number65 | 6
  Patient number66 | 6
  Patient number67 | 6
  Patient number71 | 6
  Patient number72 | 6
  Patient number74 | 6
  Patient number75 | 6
  Patient number76 | 6
  Patient number79 | 6
  Patient number80 | 6

20. Other Pre Specified Outcome: Modified OAA/S Score of Patients Receiving Intranasal Placebo at Pre-induction
Description: Modified OAA/S score of patients receiving intranasal placebo at Pre-induction.
  Modified Observer's Assessment of Alertness/Sedation Scale (Modified OAA/S score):
  6 Appears alert and awake, responds readily to name spoken in normal tone 5 Appears asleep but responds readily to name spoken in normal tone 4 Lethargic response to name spoken in normal tone 3 Responds only after name is called loudly or repeatedly 2 Responds only after mild prodding or shaking
  1 Does not respond to mild prodding or shaking 0 Does not respond to noxious stimulus
Time Frame: 1 day
Measure: Number; unit: units on a scale
Arm/Group | Placebo
Number analyzed (Participants) | 41
units on a scale
  Patient number1 | 6
  Patient number4 | 6
  Patient number8 | 5
  Patient number12 | 6
  Patient number13 | 6
  Patient number14 | 5
  Patient number15 | 6
  Patient number16 | 5
  Patient number17 | 5
  Patient number19 | 6
  Patient number20 | 6
  Patient number21 | 5
  Patient number22 | 5
  Patient number23 | 4
  Patient number26 | 6
  Patient number27 | 6
  Patient number30 | 6
  Patient number32 | 6
  Patient number34 | 6
  Patient number35 | 5
  Patient number37 | 6
  Patient number39 | 5
  Patient number41 | 5
  Patient number42 | 6
  Patient number43 | 5
  Patient number45 | 6
  Patient number47 | 6
  Patient number48 | 4
  Patient number49 | 6
  Patient number51 | 6
  Patient number54 | 4
  Patient number55 | 6
  Patient number60 | 6
  Patient number64 | 6
  Patient number68 | 6
  Patient number69 | 6
  Patient number70 | 6
  Patient number73 | 6
  Patient number77 | 6
  Patient number78 | 6
  Patient number81 | 6

21. Other Pre Specified Outcome: Modified OAA/S Score of Patients Receiving Intranasal Dexmedetomidine at Pre-induction
Description: Modified OAA/S score of patients receiving intranasal dexmedetomidine at Pre-induction.
  Modified Observer's Assessment of Alertness/Sedation Scale (Modified OAA/S score):
  6 Appears alert and awake, responds readily to name spoken in normal tone 5 Appears asleep but responds readily to name spoken in normal tone 4 Lethargic response to name spoken in normal tone 3 Responds only after name is called loudly or repeatedly 2 Responds only after mild prodding or shaking
  1 Does not respond to mild prodding or shaking 0 Does not respond to noxious stimulus
Time Frame: 1 day
Measure: Number; unit: units on a scale
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
units on a scale
  Patient number2 | 5
  Patient number3 | 5
  Patient number5 | 6
  Patient number6 | 4
  Patient number7 | 4
  Patient number9 | 5
  Patient number10 | 5
  Patient number11 | 4
  Patient number18 | 5
  Patient number24 | 5
  Patient number25 | 4
  Patient number28 | 4
  Patient number29 | 5
  Patient number31 | 6
  Patient number33 | 4
  Patient number36 | 4
  Patient number38 | 4
  Patient number40 | 4
  Patient number44 | 5
  Patient number46 | 6
  Patient number50 | 4
  Patient number52 | 4
  Patient number53 | 3
  Patient number56 | 4
  Patient number57 | 5
  Patient number58 | 4
  Patient number59 | 6
  Patient number61 | 4
  Patient number62 | 4
  Patient number63 | 4
  Patient number65 | 4
  Patient number66 | 5
  Patient number67 | 5
  Patient number71 | 4
  Patient number72 | 4
  Patient number74 | 4
  Patient number75 | 6
  Patient number76 | 5
  Patient number79 | 5
  Patient number80 | 5

22. Other Pre Specified Outcome: Modified OAA/S Score of Patients Receiving Intranasal Placebo After Extubation
Description: Modified OAA/S score of patients receiving intranasal placebo After extubation. Modified Observer's Assessment of Alertness/Sedation Scale (Modified OAA/S score) 6 Appears alert and awake, responds readily to name spoken in normal tone 5 Appears asleep but responds readily to name spoken in normal tone 4 Lethargic response to name spoken in normal tone 3 Responds only after name is called loudly or repeatedly 2 Responds only after mild prodding or shaking
  1 Does not respond to mild prodding or shaking 0 Does not respond to noxious stimulus
Time Frame: 1 day
Measure: Number; unit: units on a scale
Arm/Group | Placebo
Number analyzed (Participants) | 41
units on a scale
  Patient number1 | 4
  Patient number4 | 4
  Patient number8 | 5
  Patient number12 | 5
  Patient number13 | 4
  Patient number14 | 3
  Patient number15 | 4
  Patient number16 | 3
  Patient number17 | 6
  Patient number19 | 3
  Patient number20 | 3
  Patient number21 | 3
  Patient number22 | 4
  Patient number23 | 5
  Patient number26 | 5
  Patient number27 | 4
  Patient number30 | 5
  Patient number32 | 4
  Patient number34 | 4
  Patient number35 | 4
  Patient number37 | 3
  Patient number39 | 4
  Patient number41 | 4
  Patient number42 | 4
  Patient number43 | 4
  Patient number45 | 3
  Patient number47 | 4
  Patient number48 | 3
  Patient number49 | 3
  Patient number51 | 3
  Patient number54 | 3
  Patient number55 | 3
  Patient number60 | 4
  Patient number64 | 4
  Patient number68 | 4
  Patient number69 | 5
  Patient number70 | 5
  Patient number73 | 4
  Patient number77 | 5
  Patient number78 | 4
  Patient number81 | 6

23. Other Pre Specified Outcome: Modified OAA/S Score of Patients Receiving Intranasal Dexmedetomidine After Extubation
Description: Modified OAA/S score of patients receiving intranasal dexmedetomidine after extubation.
  Modified Observer's Assessment of Alertness/Sedation Scale (Modified OAA/S score):
  6 Appears alert and awake, responds readily to name spoken in normal tone 5 Appears asleep but responds readily to name spoken in normal tone 4 Lethargic response to name spoken in normal tone 3 Responds only after name is called loudly or repeatedly 2 Responds only after mild prodding or shaking
  1 Does not respond to mild prodding or shaking 0 Does not respond to noxious stimulus
Time Frame: 1 day
Measure: Number; unit: units on a scale
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
units on a scale
  Patient number2 | 4
  Patient number3 | 4
  Patient number5 | 4
  Patient number6 | 4
  Patient number7 | 4
  Patient number9 | 4
  Patient number10 | 4
  Patient number11 | 4
  Patient number18 | 4
  Patient number24 | 4
  Patient number25 | 4
  Patient number28 | 4
  Patient number29 | 3
  Patient number31 | 4
  Patient number33 | 4
  Patient number36 | 4
  Patient number38 | 4
  Patient number40 | 3
  Patient number44 | 4
  Patient number46 | 4
  Patient number50 | 3
  Patient number52 | 3
  Patient number53 | 3
  Patient number56 | 3
  Patient number57 | 4
  Patient number58 | 4
  Patient number59 | 3
  Patient number61 | 3
  Patient number62 | 4
  Patient number63 | 4
  Patient number65 | 4
  Patient number66 | 5
  Patient number67 | 4
  Patient number71 | 5
  Patient number72 | 5
  Patient number74 | 5
  Patient number75 | 6
  Patient number76 | 5
  Patient number79 | 3
  Patient number80 | 3

24. Other Pre Specified Outcome: Anxiety Score of Patients Receiving Intranasal Placebo Before Intranasal Drugs
Description: Anxiety score of Patients Receiving Intranasal Placebo Before Intranasal Drugs. The patients were taught to rate their anxiety levels using a 4-point anxiety score (1 = combative, 2 =anxious, 3 = calm, and 4 = amiable)
Time Frame: 1 day
Measure: Number; unit: units on a scale
Arm/Group | Placebo
Number analyzed (Participants) | 41
units on a scale
  Patient number1 | 3
  Patient number4 | 3
  Patient number8 | 3
  Patient number12 | 3
  Patient number13 | 3
  Patient number14 | 3
  Patient number15 | 2
  Patient number16 | 2
  Patient number17 | 3
  Patient number19 | 3
  Patient number20 | 3
  Patient number21 | 3
  Patient number22 | 2
  Patient number23 | 3
  Patient number26 | 2
  Patient number27 | 2
  Patient number30 | 2
  Patient number32 | 2
  Patient number34 | 3
  Patient number35 | 2
  Patient number37 | 3
  Patient number39 | 3
  Patient number41 | 2
  Patient number42 | 3
  Patient number43 | 2
  Patient number45 | 3
  Patient number47 | 3
  Patient number48 | 3
  Patient number49 | 3
  Patient number51 | 3
  Patient number54 | 2
  Patient number55 | 3
  Patient number60 | 2
  Patient number64 | 3
  Patient number68 | 2
  Patient number69 | 3
  Patient number70 | 2
  Patient number73 | 2
  Patient number77 | 2
  Patient number78 | 2
  Patient number81 | 2

25. Other Pre Specified Outcome: Anxiety Score of Patients Receiving Intranasal Dexmedetomidine Before Intranasal Drugs
Description: Anxiety score of Patients Receiving Intranasal dexmedetomidine Before Intranasal Drugs.
  The patients were taught to rate their anxiety levels using a 4-point anxiety score (1 = combative, 2 =anxious, 3 = calm, and 4 = amiable)
Time Frame: 1 day
Measure: Number; unit: units on a scale
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
units on a scale
  Patient number2 | 3
  Patient number3 | 3
  Patient number5 | 2
  Patient number6 | 2
  Patient number7 | 2
  Patient number9 | 3
  Patient number10 | 3
  Patient number11 | 3
  Patient number18 | 2
  Patient number24 | 2
  Patient number25 | 2
  Patient number28 | 3
  Patient number29 | 2
  Patient number31 | 3
  Patient number33 | 2
  Patient number36 | 3
  Patient number38 | 3
  Patient number40 | 3
  Patient number44 | 3
  Patient number46 | 3
  Patient number50 | 2
  Patient number52 | 3
  Patient number53 | 3
  Patient number56 | 2
  Patient number57 | 3
  Patient number58 | 3
  Patient number59 | 3
  Patient number61 | 3
  Patient number62 | 2
  Patient number63 | 3
  Patient number65 | 3
  Patient number66 | 3
  Patient number67 | 3
  Patient number71 | 2
  Patient number72 | 3
  Patient number74 | 3
  Patient number75 | 3
  Patient number76 | 2
  Patient number79 | 2
  Patient number80 | 2

26. Other Pre Specified Outcome: Anxiety Score of Patients Receiving Intranasal Placebo at Pre-induction
Description: Anxiety score of Patients Receiving Intranasal Placebo at Pre-induction. The patients were taught to rate their anxiety levels using a 4-point anxiety score (1 = combative, 2 =anxious, 3 = calm, and 4 = amiable)
Time Frame: 1 day
Measure: Number; unit: units on a scale
Arm/Group | Placebo
Number analyzed (Participants) | 41
units on a scale
  Patient number1 | 3
  Patient number4 | 2
  Patient number8 | 3
  Patient number12 | 3
  Patient number13 | 3
  Patient number14 | 3
  Patient number15 | 2
  Patient number16 | 3
  Patient number17 | 3
  Patient number19 | 3
  Patient number20 | 2
  Patient number21 | 3
  Patient number22 | 3
  Patient number23 | 3
  Patient number26 | 3
  Patient number27 | 3
  Patient number30 | 2
  Patient number32 | 2
  Patient number34 | 4
  Patient number35 | 4
  Patient number37 | 3
  Patient number39 | 3
  Patient number41 | 3
  Patient number42 | 2
  Patient number43 | 3
  Patient number45 | 3
  Patient number47 | 4
  Patient number48 | 4
  Patient number49 | 3
  Patient number51 | 3
  Patient number54 | 4
  Patient number55 | 3
  Patient number60 | 2
  Patient number64 | 2
  Patient number68 | 2
  Patient number69 | 3
  Patient number70 | 3
  Patient number73 | 3
  Patient number77 | 2
  Patient number78 | 2
  Patient number81 | 2

27. Other Pre Specified Outcome: Anxiety Score of Patients Receiving Intranasal Dexmedetomidine at Pre-induction
Description: Anxiety score of Patients Receiving Intranasal dexmedetomidine at Pre-induction.
  The patients were taught to rate their anxiety levels using a 4-point anxiety score (1 = combative, 2 =anxious, 3 = calm, and 4 = amiable)
Time Frame: 1 day
Measure: Number; unit: units on a scale
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
units on a scale
  Patient number2 | 3
  Patient number3 | 3
  Patient number5 | 2
  Patient number6 | 3
  Patient number7 | 3
  Patient number9 | 3
  Patient number10 | 3
  Patient number11 | 3
  Patient number18 | 3
  Patient number24 | 3
  Patient number25 | 3
  Patient number28 | 3
  Patient number29 | 3
  Patient number31 | 3
  Patient number33 | 3
  Patient number36 | 3
  Patient number38 | 4
  Patient number40 | 4
  Patient number44 | 4
  Patient number46 | 3
  Patient number50 | 4
  Patient number52 | 3
  Patient number53 | 4
  Patient number56 | 4
  Patient number57 | 4
  Patient number58 | 4
  Patient number59 | 3
  Patient number61 | 4
  Patient number62 | 4
  Patient number63 | 3
  Patient number65 | 4
  Patient number66 | 3
  Patient number67 | 3
  Patient number71 | 3
  Patient number72 | 4
  Patient number74 | 4
  Patient number75 | 3
  Patient number76 | 3
  Patient number79 | 3
  Patient number80 | 3

28. Other Pre Specified Outcome: Satisfaction Scores of Patients Receiving Intranasal Placebo
Description: Satisfaction scores of patients receiving intranasal placebo. satisfaction was assessed using a 3-point satisfaction score(1 = highly satisfactory, 2 = acceptable, and 3 = unacceptable).
Time Frame: 1 day
Measure: Number; unit: units on a scale
Arm/Group | Placebo
Number analyzed (Participants) | 41
units on a scale
  Patient number1 | 1
  Patient number4 | 1
  Patient number8 | 1
  Patient number12 | 2
  Patient number13 | 2
  Patient number14 | 1
  Patient number15 | 3
  Patient number16 | 1
  Patient number17 | 3
  Patient number19 | 2
  Patient number20 | 2
  Patient number21 | 1
  Patient number22 | 2
  Patient number23 | 1
  Patient number26 | 2
  Patient number27 | 1
  Patient number30 | 1
  Patient number32 | 2
  Patient number34 | 1
  Patient number35 | 2
  Patient number37 | 1
  Patient number39 | 2
  Patient number41 | 1
  Patient number42 | 1
  Patient number43 | 1
  Patient number45 | 1
  Patient number47 | 2
  Patient number48 | 1
  Patient number49 | 1
  Patient number51 | 2
  Patient number54 | 1
  Patient number55 | 1
  Patient number60 | 2
  Patient number64 | 1
  Patient number68 | 1
  Patient number69 | 2
  Patient number70 | 1
  Patient number73 | 2
  Patient number77 | 1
  Patient number78 | 1
  Patient number81 | 1

29. Other Pre Specified Outcome: Satisfaction Scores of Patients Receiving Intranasal Dexmedetomidine
Description: Satisfaction scores of patients receiving intranasal dexmedetomidine. Satisfaction used a 3-point satisfaction score(1 = highly satisfactory, 2 = acceptable, and 3 = unacceptable).
Time Frame: 1 day
Measure: Number; unit: units on a scale
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
units on a scale
  Patient number2 | 1
  Patient number3 | 1
  Patient number5 | 1
  Patient number6 | 1
  Patient number7 | 1
  Patient number9 | 1
  Patient number10 | 1
  Patient number11 | 2
  Patient number18 | 1
  Patient number24 | 1
  Patient number25 | 1
  Patient number28 | 1
  Patient number29 | 1
  Patient number31 | 2
  Patient number33 | 1
  Patient number36 | 1
  Patient number38 | 1
  Patient number40 | 1
  Patient number44 | 2
  Patient number46 | 1
  Patient number50 | 1
  Patient number52 | 1
  Patient number53 | 1
  Patient number56 | 1
  Patient number57 | 1
  Patient number58 | 2
  Patient number59 | 1
  Patient number61 | 1
  Patient number62 | 1
  Patient number63 | 1
  Patient number65 | 1
  Patient number66 | 1
  Patient number67 | 1
  Patient number71 | 1
  Patient number72 | 1
  Patient number74 | 1
  Patient number75 | 1
  Patient number76 | 1
  Patient number79 | 2
  Patient number80 | 2

30. Secondary Outcome: Number of Participants With Anxiety Score >2
Description: satisfaction using a 3-point satisfaction score (1 = highly satisfactory, 2 = acceptable, and 3 = unacceptable) anxiety levels using a 4-point anxiety score (1 = combative, 2 = anxious, 3 = calm, and 4 = amiable) were collected before intranasal drugs and at pre-induction.
  Anxiety score >2 was considered to be better for the patient.
Time Frame: 1 day
Measure: Number; unit: participant
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 40 | 41
participant
  Before intranasal drugs | 25 | 23
  Pre-induction | 39 | 29

31. Other Pre Specified Outcome: Time to Spontaneous Breathing of Patients Receiving Intranasal Placebo
Description: Time to spontaneous breathing of patients receiving intranasal placebo. The time elapsed between stopping anesthetic infusions and adequate ventilation
Time Frame: 1 day
Measure: Number; unit: minutes
Arm/Group | Placebo
Number analyzed (Participants) | 41
minutes
  Patient number1 | 5
  Patient number4 | 5
  Patient number8 | 7
  Patient number12 | 7
  Patient number13 | 9
  Patient number14 | 7
  Patient number15 | 11
  Patient number16 | 10
  Patient number17 | 9
  Patient number19 | 10
  Patient number20 | 5
  Patient number21 | 9
  Patient number22 | 9
  Patient number23 | 8
  Patient number26 | 15
  Patient number27 | 8
  Patient number30 | 13
  Patient number32 | 8
  Patient number34 | 7
  Patient number35 | 8
  Patient number37 | 8
  Patient number39 | 9
  Patient number41 | 8
  Patient number42 | 8
  Patient number43 | 7
  Patient number45 | 6
  Patient number47 | 7
  Patient number48 | 6
  Patient number49 | 4
  Patient number51 | 8
  Patient number54 | 3
  Patient number55 | 15
  Patient number60 | 5
  Patient number64 | 11
  Patient number68 | 7
  Patient number69 | 6
  Patient number70 | 4
  Patient number73 | 8
  Patient number77 | 8
  Patient number78 | 8
  Patient number81 | 7

32. Other Pre Specified Outcome: Time to Spontaneous Breathing of Patients Receiving Intranasal Dexmedetomidine
Description: Time to spontaneous breathing of patients receiving intranasal dexmedetomidine. The time elapsed between stopping anesthetic infusions and adequate ventilation
Time Frame: 1 day
Measure: Number; unit: minutes
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
minutes
  Patient number2 | 6
  Patient number3 | 5
  Patient number5 | 8
  Patient number6 | 6
  Patient number7 | 8
  Patient number9 | 8
  Patient number10 | 6
  Patient number11 | 8
  Patient number18 | 7
  Patient number24 | 18
  Patient number25 | 10
  Patient number28 | 5
  Patient number29 | 8
  Patient number31 | 10
  Patient number33 | 9
  Patient number36 | 6
  Patient number38 | 8
  Patient number40 | 8
  Patient number44 | 10
  Patient number46 | 7
  Patient number50 | 7
  Patient number52 | 7
  Patient number53 | 5
  Patient number56 | 7
  Patient number57 | 8
  Patient number58 | 6
  Patient number59 | 9
  Patient number61 | 6
  Patient number62 | 7
  Patient number63 | 13
  Patient number65 | 10
  Patient number66 | 7
  Patient number67 | 11
  Patient number71 | 6
  Patient number72 | 8
  Patient number74 | 8
  Patient number75 | 5
  Patient number76 | 11
  Patient number79 | 7
  Patient number80 | 20

33. Other Pre Specified Outcome: Time to Consciousness of Patients Receiving Intranasal Placebo
Description: Time to consciousness of patients receiving intranasal placebo. The time elapsed between stopping anesthetic infusions and consciousness.
Time Frame: 1 day
Measure: Number; unit: minutes
Arm/Group | Placebo
Number analyzed (Participants) | 41
minutes
  Patient number1 | 9
  Patient number4 | 10
  Patient number8 | 9
  Patient number12 | 8
  Patient number13 | 14
  Patient number14 | 12
  Patient number15 | 29
  Patient number16 | 15
  Patient number17 | 17
  Patient number19 | 19
  Patient number20 | 20
  Patient number21 | 15
  Patient number22 | 12
  Patient number23 | 11
  Patient number26 | 16
  Patient number27 | 17
  Patient number30 | 15
  Patient number32 | 14
  Patient number34 | 16
  Patient number35 | 14
  Patient number37 | 12
  Patient number39 | 15
  Patient number41 | 16
  Patient number42 | 14
  Patient number43 | 15
  Patient number45 | 13
  Patient number47 | 10
  Patient number48 | 8
  Patient number49 | 14
  Patient number51 | 16
  Patient number54 | 5
  Patient number55 | 26
  Patient number60 | 13
  Patient number64 | 14
  Patient number68 | 11
  Patient number69 | 12
  Patient number70 | 14
  Patient number73 | 21
  Patient number77 | 11
  Patient number78 | 14
  Patient number81 | 41

34. Other Pre Specified Outcome: Time to Consciousness of Patients Receiving Intranasal Dexmedetomidine
Description: Time to consciousness of patients receiving intranasal dexmedetomidine. The time elapsed between stopping anesthetic infusions and consciousness.
Time Frame: 1 day
Measure: Number; unit: minutes
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
minutes
  Patient number2 | 11
  Patient number3 | 14
  Patient number5 | 16
  Patient number6 | 11
  Patient number7 | 18
  Patient number9 | 13
  Patient number10 | 15
  Patient number11 | 11
  Patient number18 | 12
  Patient number24 | 23
  Patient number25 | 14
  Patient number28 | 12
  Patient number29 | 31
  Patient number31 | 16
  Patient number33 | 19
  Patient number36 | 12
  Patient number38 | 18
  Patient number40 | 16
  Patient number44 | 41
  Patient number46 | 14
  Patient number50 | 14
  Patient number52 | 10
  Patient number53 | 10
  Patient number56 | 19
  Patient number57 | 17
  Patient number58 | 17
  Patient number59 | 16
  Patient number61 | 20
  Patient number62 | 19
  Patient number63 | 24
  Patient number65 | 19
  Patient number66 | 12
  Patient number67 | 18
  Patient number71 | 10
  Patient number72 | 11
  Patient number74 | 10
  Patient number75 | 14
  Patient number76 | 13
  Patient number79 | 14
  Patient number80 | 25

35. Other Pre Specified Outcome: Time to Extubation of Patients Receiving Intranasal Placebo
Description: Time to extubation of patients receiving intranasal placebo. The time elapsed between stopping anesthetic infusions and extubation
Time Frame: 1 day
Measure: Number; unit: minutes
Arm/Group | Placebo
Number analyzed (Participants) | 41
minutes
  Patient number1 | 11
  Patient number4 | 12
  Patient number8 | 10
  Patient number12 | 10
  Patient number13 | 16
  Patient number14 | 14
  Patient number15 | 35
  Patient number16 | 17
  Patient number17 | 19
  Patient number19 | 21
  Patient number20 | 22
  Patient number21 | 17
  Patient number22 | 14
  Patient number23 | 12
  Patient number26 | 16
  Patient number27 | 17
  Patient number30 | 18
  Patient number32 | 16
  Patient number34 | 19
  Patient number35 | 18
  Patient number37 | 14
  Patient number39 | 17
  Patient number41 | 18
  Patient number42 | 16
  Patient number43 | 16
  Patient number45 | 18
  Patient number47 | 12
  Patient number48 | 9
  Patient number49 | 16
  Patient number51 | 20
  Patient number54 | 8
  Patient number55 | 29
  Patient number60 | 15
  Patient number64 | 15
  Patient number68 | 13
  Patient number69 | 14
  Patient number70 | 16
  Patient number73 | 26
  Patient number77 | 13
  Patient number78 | 17
  Patient number81 | 46

36. Other Pre Specified Outcome: Time to Extubation of Patients Receiving Intranasal Dexmedetomidine
Description: Time to extubation of patients receiving intranasal dexmedetomidine. The time elapsed between stopping anesthetic infusions and extubation
Time Frame: 1 day
Measure: Number; unit: minutes
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
minutes
  Patient number2 | 12
  Patient number3 | 15
  Patient number5 | 18
  Patient number6 | 13
  Patient number7 | 20
  Patient number9 | 15
  Patient number10 | 16
  Patient number11 | 13
  Patient number18 | 14
  Patient number24 | 25
  Patient number25 | 16
  Patient number28 | 14
  Patient number29 | 36
  Patient number31 | 18
  Patient number33 | 22
  Patient number36 | 17
  Patient number38 | 21
  Patient number40 | 18
  Patient number44 | 48
  Patient number46 | 16
  Patient number50 | 16
  Patient number52 | 11
  Patient number53 | 11
  Patient number56 | 21
  Patient number57 | 17
  Patient number58 | 19
  Patient number59 | 19
  Patient number61 | 23
  Patient number62 | 22
  Patient number63 | 26
  Patient number65 | 23
  Patient number66 | 14
  Patient number67 | 22
  Patient number71 | 11
  Patient number72 | 12
  Patient number74 | 11
  Patient number75 | 15
  Patient number76 | 15
  Patient number79 | 16
  Patient number80 | 30

37. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Propofol After Intranasal Placebo at Tracheal Intubation
Description: Predicted effect-site concentrations of propofol after intranasal placebo at tracheal intubation.
  Propofol was infused intraoperatively to a target-controlled infusion (TCI) plasma concentration of 2.5μg∙ml-1 using DiprifusorTM software. The infusion rate was adjusted via plasma concentration increments of 0.5 μg∙ml-1 at 2-min intervals to maintain the Narcotrend index between 'D0' and 'E1' until the end of surgery.
Time Frame: 1 day
Measure: Number; unit: µg/ml
Arm/Group | Placebo
Number analyzed (Participants) | 41
µg/ml
  Patient number1 | 2.1
  Patient number4 | 2.5
  Patient number8 | 1.4
  Patient number12 | 1.4
  Patient number13 | 1.1
  Patient number14 | 3.6
  Patient number15 | 1.4
  Patient number16 | 2.4
  Patient number17 | 2.6
  Patient number19 | 4.3
  Patient number20 | 2.1
  Patient number21 | 3
  Patient number22 | 1.9
  Patient number23 | 1
  Patient number26 | 3.3
  Patient number27 | 2.5
  Patient number30 | 3.3
  Patient number32 | 3.8
  Patient number34 | 2.2
  Patient number35 | 1
  Patient number37 | 2.1
  Patient number39 | 3.3
  Patient number41 | 3.5
  Patient number42 | 2.1
  Patient number43 | 2.6
  Patient number45 | 3.2
  Patient number47 | 2.4
  Patient number48 | 2.9
  Patient number49 | 2.2
  Patient number51 | 1.7
  Patient number54 | 1.5
  Patient number55 | 2.2
  Patient number60 | 2.7
  Patient number64 | 2.4
  Patient number68 | 2.5
  Patient number69 | 2.3
  Patient number70 | 1.2
  Patient number73 | 1.7
  Patient number77 | 1.7
  Patient number78 | 1.7
  Patient number81 | 2.3

38. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Propofol After Intranasal Dexmedetomidine at Tracheal Intubation
Description: Predicted effect-site concentrations of propofol after intranasal dexmedetomidine at tracheal intubation.
  Propofol was infused intraoperatively to a TCI plasma concentration of 2.5μg∙ml-1 using DiprifusorTM software. The infusion rate was adjusted via plasma concentration increments of 0.5 μg∙ml-1 at 2-min intervals to maintain the Narcotrend index between 'D0' and 'E1' until the end of surgery.
Time Frame: 1 day
Measure: Number; unit: µg/ml
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
µg/ml
  Patient number2 | 1.4
  Patient number3 | 1.7
  Patient number5 | 4
  Patient number6 | 2.9
  Patient number7 | 0.7
  Patient number9 | 2.7
  Patient number10 | 1.8
  Patient number11 | 1.6
  Patient number18 | 1.8
  Patient number24 | 2
  Patient number25 | 0.9
  Patient number28 | 2
  Patient number29 | 2.5
  Patient number31 | 1.6
  Patient number33 | 2.8
  Patient number36 | 1.9
  Patient number38 | 1.8
  Patient number40 | 2.2
  Patient number44 | 1.8
  Patient number46 | 3.2
  Patient number50 | 1.1
  Patient number52 | 1.4
  Patient number53 | 2.3
  Patient number56 | 1.7
  Patient number57 | 2
  Patient number58 | 1.6
  Patient number59 | 2.7
  Patient number61 | 1.6
  Patient number62 | 1.5
  Patient number63 | 2.1
  Patient number65 | 1.3
  Patient number66 | 2.1
  Patient number67 | 2.9
  Patient number71 | 1.6
  Patient number72 | 3
  Patient number74 | 2
  Patient number75 | 2.3
  Patient number76 | 4.1
  Patient number79 | 2.1
  Patient number80 | 1.6

39. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Propofol After Intranasal Placebo Before Inserting Operative Laryngoscope
Description: Predicted effect-site concentrations of propofol after intranasal placebo before inserting operative laryngoscope.
  Propofol was infused intraoperatively to a TCI plasma concentration of 2.5μg∙ml-1 using DiprifusorTM software. The infusion rate was adjusted via plasma concentration increments of 0.5 μg∙ml-1 at 2-min intervals to maintain the Narcotrend index between 'D0' and 'E1' until the end of surgery.
Time Frame: 1 day
Measure: Number; unit: µg/ml
Arm/Group | Placebo
Number analyzed (Participants) | 41
µg/ml
  Patient number1 | 3
  Patient number4 | 3.5
  Patient number8 | 3
  Patient number12 | 3
  Patient number13 | 2.5
  Patient number14 | 4.9
  Patient number15 | 3.4
  Patient number16 | 3.5
  Patient number17 | 4
  Patient number19 | 5
  Patient number20 | 3.5
  Patient number21 | 4.3
  Patient number22 | 3.8
  Patient number23 | 2.5
  Patient number26 | 4.5
  Patient number27 | 3.4
  Patient number30 | 4.5
  Patient number32 | 4.9
  Patient number34 | 3.9
  Patient number35 | 2.9
  Patient number37 | 4.4
  Patient number39 | 4
  Patient number41 | 4.5
  Patient number42 | 3.5
  Patient number43 | 4
  Patient number45 | 3.9
  Patient number47 | 3.9
  Patient number48 | 4
  Patient number49 | 3.5
  Patient number51 | 3
  Patient number54 | 3
  Patient number55 | 3.5
  Patient number60 | 4.5
  Patient number64 | 3.9
  Patient number68 | 3.3
  Patient number69 | 3.4
  Patient number70 | 3
  Patient number73 | 3.4
  Patient number77 | 2.9
  Patient number78 | 3.5
  Patient number81 | 3.7

40. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Propofol After Intranasal Dexmedetomidine Before Inserting Operative Laryngoscope
Description: Predicted effect-site concentrations of propofol after intranasal dexmedetomidine before inserting operative laryngoscope.
  Propofol was infused intraoperatively to a TCI plasma concentration of 2.5μg∙ml-1 using DiprifusorTM software. The infusion rate was adjusted via plasma concentration increments of 0.5 μg∙ml-1 at 2-min intervals to maintain the Narcotrend index between 'D0' and 'E1' until the end of surgery.
Time Frame: 1 day
Measure: Number; unit: µg/ml
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
µg/ml
  Patient number2 | 3
  Patient number3 | 2.8
  Patient number5 | 4.9
  Patient number6 | 4
  Patient number7 | 2.4
  Patient number9 | 4
  Patient number10 | 2.9
  Patient number11 | 2.9
  Patient number18 | 2.7
  Patient number24 | 3.3
  Patient number25 | 3
  Patient number28 | 3
  Patient number29 | 3.5
  Patient number31 | 3
  Patient number33 | 3.9
  Patient number36 | 3.5
  Patient number38 | 3.4
  Patient number40 | 3.5
  Patient number44 | 2.9
  Patient number46 | 4.4
  Patient number50 | 3
  Patient number52 | 2.9
  Patient number53 | 3.3
  Patient number56 | 2.9
  Patient number57 | 3.4
  Patient number58 | 3
  Patient number59 | 4
  Patient number61 | 3
  Patient number62 | 3
  Patient number63 | 3.5
  Patient number65 | 3.5
  Patient number66 | 3.5
  Patient number67 | 3.9
  Patient number71 | 3
  Patient number72 | 4.2
  Patient number74 | 3.5
  Patient number75 | 3.5
  Patient number76 | 4.9
  Patient number79 | 3.4
  Patient number80 | 3

41. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Propofol After Intranasal Placebo on Removal of Operative Laryngoscope
Description: Predicted effect-site concentrations of propofol after intranasal placebo on removal of operative laryngoscope.
  Propofol was infused intraoperatively to a TCI plasma concentration of 2.5μg∙ml-1 using DiprifusorTM software. The infusion rate was adjusted via plasma concentration increments of 0.5 μg∙ml-1 at 2-min intervals to maintain the Narcotrend index between 'D0' and 'E1' until the end of surgery.
Time Frame: 1 day
Measure: Number; unit: µg/ml
Arm/Group | Placebo
Number analyzed (Participants) | 41
µg/ml
  Patient number1 | 3
  Patient number4 | 3.5
  Patient number8 | 3
  Patient number12 | 3
  Patient number13 | 2.5
  Patient number14 | 4.5
  Patient number15 | 3.5
  Patient number16 | 3.5
  Patient number17 | 4
  Patient number19 | 4.5
  Patient number20 | 3.5
  Patient number21 | 4.5
  Patient number22 | 4
  Patient number23 | 2.5
  Patient number26 | 4
  Patient number27 | 3
  Patient number30 | 4.5
  Patient number32 | 5
  Patient number34 | 4
  Patient number35 | 3
  Patient number37 | 4.5
  Patient number39 | 4
  Patient number41 | 4.5
  Patient number42 | 3.5
  Patient number43 | 4
  Patient number45 | 4
  Patient number47 | 4
  Patient number48 | 4
  Patient number49 | 3.5
  Patient number51 | 3
  Patient number54 | 3
  Patient number55 | 3.5
  Patient number60 | 4.5
  Patient number64 | 4
  Patient number68 | 3.5
  Patient number69 | 3.5
  Patient number70 | 3
  Patient number73 | 3.5
  Patient number77 | 3
  Patient number78 | 3.5
  Patient number81 | 3.6

42. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Propofol After Intranasal Dexmedetomidine on Removal of Operative Laryngoscope
Description: Predicted effect-site concentrations of propofol after intranasal dexmedetomidine on removal of operative laryngoscope.
  Propofol was infused intraoperatively to a TCI plasma concentration of 2.5μg∙ml-1 using DiprifusorTM software. The infusion rate was adjusted via plasma concentration increments of 0.5 μg∙ml-1 at 2-min intervals to maintain the Narcotrend index between 'D0' and 'E1' until the end of surgery.
Time Frame: 1 day
Measure: Number; unit: µg/ml
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
µg/ml
  Patient number2 | 3
  Patient number3 | 3
  Patient number5 | 5
  Patient number6 | 4
  Patient number7 | 2.5
  Patient number9 | 4
  Patient number10 | 3
  Patient number11 | 3
  Patient number18 | 3
  Patient number24 | 3.5
  Patient number25 | 3
  Patient number28 | 3
  Patient number29 | 4
  Patient number31 | 3
  Patient number33 | 4
  Patient number36 | 4
  Patient number38 | 3.5
  Patient number40 | 3.5
  Patient number44 | 3
  Patient number46 | 4.5
  Patient number50 | 3
  Patient number52 | 3
  Patient number53 | 4
  Patient number56 | 3
  Patient number57 | 3.5
  Patient number58 | 3
  Patient number59 | 4
  Patient number61 | 3
  Patient number62 | 3
  Patient number63 | 3.5
  Patient number65 | 3
  Patient number66 | 3.5
  Patient number67 | 4
  Patient number71 | 3
  Patient number72 | 4.5
  Patient number74 | 3.5
  Patient number75 | 3.5
  Patient number76 | 5
  Patient number79 | 3
  Patient number80 | 3

43. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Propofol After Intranasal Placebo at Return of Spontaneous Breathing
Description: Predicted effect-site concentrations of propofol after intranasal placebo at return of spontaneous breathing.
  Propofol was infused intraoperatively to a TCI plasma concentration of 2.5μg∙ml-1 using DiprifusorTM software. The infusion rate was adjusted via plasma concentration increments of 0.5 μg∙ml-1 at 2-min intervals to maintain the Narcotrend index between 'D0' and 'E1' until the end of surgery.
Time Frame: 1 day
Measure: Number; unit: ug/ml
Arm/Group | Placebo
Number analyzed (Participants) | 41
ug/ml
  Patient number1 | 2.1
  Patient number4 | 2.3
  Patient number8 | 1.7
  Patient number12 | 1.7
  Patient number13 | 1
  Patient number14 | 2.5
  Patient number15 | 1.2
  Patient number16 | 1.3
  Patient number17 | 1.7
  Patient number19 | 1.9
  Patient number20 | 2.3
  Patient number21 | 2.1
  Patient number22 | 0.7
  Patient number23 | 1.1
  Patient number26 | 1.9
  Patient number27 | 1.8
  Patient number30 | 1.3
  Patient number32 | 2.5
  Patient number34 | 2.1
  Patient number35 | 1.5
  Patient number37 | 2.3
  Patient number39 | 1.7
  Patient number41 | 2.3
  Patient number42 | 1.7
  Patient number43 | 2.1
  Patient number45 | 2.3
  Patient number47 | 2.1
  Patient number48 | 2.3
  Patient number49 | 2.5
  Patient number51 | 1.5
  Patient number54 | 2.5
  Patient number55 | 0.9
  Patient number60 | 2.9
  Patient number64 | 1.3
  Patient number68 | 1.9
  Patient number69 | 2.1
  Patient number70 | 2.3
  Patient number73 | 1.7
  Patient number77 | 1.5
  Patient number78 | 1.9
  Patient number81 | 1.9

44. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Propofol After Intranasal Dexmedetomidine at Return of Spontaneous Breathing
Description: Predicted effect-site concentrations of propofol after intranasal dexmedetomidine at return of spontaneous breathing.
  Propofol was infused intraoperatively to a TCI plasma concentration of 2.5μg∙ml-1 using DiprifusorTM software. The infusion rate was adjusted via plasma concentration increments of 0.5 μg∙ml-1 at 2-min intervals to maintain the Narcotrend index between 'D0' and 'E1' until the end of surgery.
Time Frame: 1 day
Measure: Number; unit: µg/ml
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
µg/ml
  Patient number2 | 1.9
  Patient number3 | 2.1
  Patient number5 | 1.7
  Patient number6 | 2.3
  Patient number7 | 1.1
  Patient number9 | 1.9
  Patient number10 | 1.9
  Patient number11 | 1.5
  Patient number18 | 1.7
  Patient number24 | 0.7
  Patient number25 | 1.2
  Patient number28 | 2.1
  Patient number29 | 1.9
  Patient number31 | 1.2
  Patient number33 | 1.7
  Patient number36 | 2.3
  Patient number38 | 1.7
  Patient number40 | 1.7
  Patient number44 | 1.2
  Patient number46 | 2.5
  Patient number50 | 1.7
  Patient number52 | 1.7
  Patient number53 | 2.5
  Patient number56 | 1.7
  Patient number57 | 1.7
  Patient number58 | 1.9
  Patient number59 | 1.7
  Patient number61 | 1.9
  Patient number62 | 1.7
  Patient number63 | 1
  Patient number65 | 1.2
  Patient number66 | 1.9
  Patient number67 | 1.3
  Patient number71 | 1.9
  Patient number72 | 2.3
  Patient number74 | 1.7
  Patient number75 | 2.3
  Patient number76 | 1.9
  Patient number79 | 1.7
  Patient number80 | 0.6

45. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Propofol After Intranasal Placebo at Emergence
Description: Predicted effect-site concentrations of propofol after intranasal placebo at emergence.
  Propofol was infused intraoperatively to a TCI plasma concentration of 2.5μg∙ml-1 using DiprifusorTM software. The infusion rate was adjusted via plasma concentration increments of 0.5 μg∙ml-1 at 2-min intervals to maintain the Narcotrend index between 'D0' and 'E1' until the end of surgery.
Time Frame: 1 day
Measure: Number; unit: µg/ml
Arm/Group | Placebo
Number analyzed (Participants) | 41
µg/ml
  Patient number1 | 1.3
  Patient number4 | 1.3
  Patient number8 | 1.3
  Patient number12 | 1.5
  Patient number13 | 0.7
  Patient number14 | 1.5
  Patient number15 | 0.5
  Patient number16 | 0.9
  Patient number17 | 0.8
  Patient number19 | 0.8
  Patient number20 | 0.6
  Patient number21 | 1.1
  Patient number22 | 1.2
  Patient number23 | 0.9
  Patient number26 | 1
  Patient number27 | 1
  Patient number30 | 1.1
  Patient number32 | 1.3
  Patient number34 | 0.9
  Patient number35 | 0.9
  Patient number37 | 1.5
  Patient number39 | 0.9
  Patient number41 | 1
  Patient number42 | 0.9
  Patient number43 | 0.9
  Patient number45 | 1.1
  Patient number47 | 1.5
  Patient number48 | 1.9
  Patient number49 | 0.9
  Patient number51 | 0.7
  Patient number54 | 2.1
  Patient number55 | 0.5
  Patient number60 | 1.3
  Patient number64 | 1
  Patient number68 | 1.2
  Patient number69 | 1.1
  Patient number70 | 0.9
  Patient number73 | 0.6
  Patient number77 | 1.1
  Patient number78 | 0.2
  Patient number81 | 1.1

46. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Propofol After Intranasal Dexmedetomidine at Emergence
Description: Predicted effect-site concentrations of propofol after intranasal dexmedetomidine at emergence.
  Propofol was infused intraoperatively to a TCI plasma concentration of 2.5μg∙ml-1 using DiprifusorTM software. The infusion rate was adjusted via plasma concentration increments of 0.5 μg∙ml-1 at 2-min intervals to maintain the Narcotrend index between 'D0' and 'E1' until the end of surgery.
Time Frame: 1 day
Measure: Number; unit: µg/ml
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
µg/ml
  Patient number2 | 1.1
  Patient number3 | 0.9
  Patient number5 | 0.8
  Patient number6 | 1.3
  Patient number7 | 0.8
  Patient number9 | 1.1
  Patient number10 | 0.8
  Patient number11 | 1.1
  Patient number18 | 1
  Patient number24 | 0.6
  Patient number25 | 0.9
  Patient number28 | 1
  Patient number29 | 0.5
  Patient number31 | 0.7
  Patient number33 | 0.7
  Patient number36 | 1.2
  Patient number38 | 0.7
  Patient number40 | 0.8
  Patient number44 | 0.2
  Patient number46 | 1.2
  Patient number50 | 0.9
  Patient number52 | 1.2
  Patient number53 | 1.5
  Patient number56 | 0.6
  Patient number57 | 0.9
  Patient number58 | 0.7
  Patient number59 | 0.9
  Patient number61 | 0.6
  Patient number62 | 0.6
  Patient number63 | 0.5
  Patient number65 | 0.6
  Patient number66 | 1.1
  Patient number67 | 0.7
  Patient number71 | 1.2
  Patient number72 | 1.7
  Patient number74 | 1.3
  Patient number75 | 0.9
  Patient number76 | 1.5
  Patient number79 | 0.9
  Patient number80 | 0.5

47. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Propofol After Intranasal Placebo at Extubation
Description: Predicted effect-site concentrations of propofol after intranasal placebo at extubation.
  Propofol was infused intraoperatively to a TCI plasma concentration of 2.5μg∙ml-1 using DiprifusorTM software. The infusion rate was adjusted via plasma concentration increments of 0.5 μg∙ml-1 at 2-min intervals to maintain the Narcotrend index between 'D0' and 'E1' until the end of surgery.
Time Frame: 1 day
Measure: Number; unit: µg/ml
Arm/Group | Placebo
Number analyzed (Participants) | 41
µg/ml
  Patient number1 | 1.1
  Patient number4 | 1.1
  Patient number8 | 1.2
  Patient number12 | 1.2
  Patient number13 | 0.6
  Patient number14 | 1.2
  Patient number15 | 0.4
  Patient number16 | 0.7
  Patient number17 | 0.7
  Patient number19 | 0.7
  Patient number20 | 0.6
  Patient number21 | 0.9
  Patient number22 | 1
  Patient number23 | 0.8
  Patient number26 | 0.9
  Patient number27 | 0.8
  Patient number30 | 0.9
  Patient number32 | 1.1
  Patient number34 | 0.7
  Patient number35 | 0.7
  Patient number37 | 1.2
  Patient number39 | 0.8
  Patient number41 | 0.9
  Patient number42 | 0.8
  Patient number43 | 0.9
  Patient number45 | 0.7
  Patient number47 | 1.2
  Patient number48 | 1.7
  Patient number49 | 0.8
  Patient number51 | 0.6
  Patient number54 | 1.5
  Patient number55 | 0.4
  Patient number60 | 1.1
  Patient number64 | 0.9
  Patient number68 | 1
  Patient number69 | 0.9
  Patient number70 | 0.7
  Patient number73 | 0.5
  Patient number77 | 0.9
  Patient number78 | 0.2
  Patient number81 | 0.9

48. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Propofol After Intranasal Dexmedetomidine at Extubation
Description: Predicted effect-site concentrations of propofol after intranasal dexmedetomidine at extubation.
  Propofol was infused intraoperatively to a TCI plasma concentration of 2.5μg∙ml-1 using DiprifusorTM software. The infusion rate was adjusted via plasma concentration increments of 0.5 μg∙ml-1 at 2-min intervals to maintain the Narcotrend index between 'D0' and 'E1' until the end of surgery.
Time Frame: 1 day
Measure: Number; unit: µg/ml
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
µg/ml
  Patient number2 | 1
  Patient number3 | 0.8
  Patient number5 | 0.7
  Patient number6 | 1.1
  Patient number7 | 0.5
  Patient number9 | 0.9
  Patient number10 | 0.7
  Patient number11 | 0.9
  Patient number18 | 0.9
  Patient number24 | 0.5
  Patient number25 | 0.7
  Patient number28 | 0.9
  Patient number29 | 0.5
  Patient number31 | 0.7
  Patient number33 | 0.6
  Patient number36 | 0.8
  Patient number38 | 0.6
  Patient number40 | 0.7
  Patient number44 | 0.2
  Patient number46 | 1.1
  Patient number50 | 0.7
  Patient number52 | 1.1
  Patient number53 | 1.3
  Patient number56 | 0.6
  Patient number57 | 0.8
  Patient number58 | 0.6
  Patient number59 | 0.7
  Patient number61 | 0.5
  Patient number62 | 0.6
  Patient number63 | 0.5
  Patient number65 | 0.5
  Patient number66 | 0.9
  Patient number67 | 0.6
  Patient number71 | 1.1
  Patient number72 | 1.5
  Patient number74 | 1.2
  Patient number75 | 0.9
  Patient number76 | 1.2
  Patient number79 | 0.8
  Patient number80 | 0.4

49. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Remifentanil After Intranasal Placebo at Tracheal Intubation
Description: Predicted effect-site concentrations of remifentanil after intranasal placebo at tracheal intubation.
  Remifentanil was infused to achieve a TCI plasma concentration of 3.0 ng∙ml-1 using the Minto pharmacokinetic model 24 and then adjusted to maintain the systolic blood pressure (SBP) at 25% of the pre-operative value and the HR at less than 90 bpm. To maintain a neuromuscular blockade, 0.15 mg∙kg-1 increments of rocuronium were infused upon observation of the first twitch in a train-of-four response with the nerve stimulator
Time Frame: 1 day
Measure: Number; unit: ng/ml
Arm/Group | Placebo
Number analyzed (Participants) | 41
ng/ml
  Patient number1 | 3
  Patient number4 | 3
  Patient number8 | 3
  Patient number12 | 3
  Patient number13 | 3
  Patient number14 | 3
  Patient number15 | 3
  Patient number16 | 3
  Patient number17 | 3
  Patient number19 | 3
  Patient number20 | 3
  Patient number21 | 3
  Patient number22 | 3
  Patient number23 | 3
  Patient number26 | 3
  Patient number27 | 3
  Patient number30 | 3
  Patient number32 | 3
  Patient number34 | 3
  Patient number35 | 3
  Patient number37 | 3
  Patient number39 | 3
  Patient number41 | 3
  Patient number42 | 3
  Patient number43 | 3
  Patient number45 | 3
  Patient number47 | 3
  Patient number48 | 3
  Patient number49 | 3
  Patient number51 | 3
  Patient number54 | 3
  Patient number55 | 3
  Patient number60 | 3
  Patient number64 | 3
  Patient number68 | 3
  Patient number69 | 3
  Patient number70 | 3
  Patient number73 | 3
  Patient number77 | 3
  Patient number81 | 3
  Patient number78 | 3

50. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Remifentanil After Intranasal Dexmedetomidine at Tracheal Intubation
Description: Predicted effect-site concentrations of remifentanil after intranasal dexmedetomidine at tracheal intubation.
  Remifentanil was infused to achieve a TCI plasma concentration of 3.0 ng∙ml-1 using the Minto pharmacokinetic model 24 and then adjusted to maintain the systolic blood pressure (SBP) at 25% of the pre-operative value and the HR at less than 90 bpm. To maintain a neuromuscular blockade, 0.15 mg∙kg-1 increments of rocuronium were infused upon observation of the first twitch in a train-of-four response with the nerve stimulator
Time Frame: 1 day
Measure: Number; unit: ng/ml
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
ng/ml
  Patient number2 | 3
  Patient number3 | 3
  Patient number5 | 3
  Patient number6 | 3
  Patient number7 | 3
  Patient number9 | 3
  Patient number10 | 3
  Patient number11 | 3
  Patient number18 | 3
  Patient number24 | 3
  Patient number25 | 3
  Patient number28 | 3
  Patient number29 | 3
  Patient number31 | 3
  Patient number33 | 3
  Patient number36 | 3
  Patient number38 | 3
  Patient number40 | 3
  Patient number44 | 3
  Patient number46 | 3
  Patient number50 | 3
  Patient number52 | 3
  Patient number53 | 3
  Patient number56 | 3
  Patient number57 | 3
  Patient number58 | 3
  Patient number59 | 3
  Patient number61 | 3
  Patient number62 | 3
  Patient number63 | 3
  Patient number65 | 3
  Patient number66 | 3
  Patient number67 | 3
  Patient number71 | 3
  Patient number72 | 3
  Patient number74 | 3
  Patient number75 | 3
  Patient number76 | 3
  Patient number79 | 3
  Patient number80 | 3

51. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Remifentanil After Intranasal Placebo Before Inserting Operative Laryngoscope
Description: Predicted effect-site concentrations of remifentanil after intranasal placebo before inserting operative laryngoscope.
  Remifentanil was infused to achieve a TCI plasma concentration of 3.0 ng∙ml-1 using the Minto pharmacokinetic model 24 and then adjusted to maintain the systolic blood pressure (SBP) at 25% of the pre-operative value and the HR at less than 90 bpm. To maintain a neuromuscular blockade, 0.15 mg∙kg-1 increments of rocuronium were infused upon observation of the first twitch in a train-of-four response with the nerve stimulator
Time Frame: 1 day
Measure: Number; unit: ng/ml
Arm/Group | Placebo
Number analyzed (Participants) | 41
ng/ml
  Patient number1 | 2
  Patient number4 | 2.5
  Patient number8 | 2.5
  Patient number12 | 3.5
  Patient number13 | 2
  Patient number14 | 3
  Patient number15 | 2
  Patient number16 | 3
  Patient number17 | 2
  Patient number19 | 2
  Patient number20 | 2
  Patient number21 | 2
  Patient number22 | 2
  Patient number23 | 2
  Patient number26 | 3
  Patient number27 | 2
  Patient number30 | 2
  Patient number32 | 2.5
  Patient number34 | 2
  Patient number35 | 2
  Patient number37 | 2.5
  Patient number39 | 3
  Patient number41 | 2.5
  Patient number42 | 2.5
  Patient number43 | 2
  Patient number45 | 3
  Patient number47 | 3
  Patient number48 | 2
  Patient number49 | 2.5
  Patient number51 | 2
  Patient number54 | 2.5
  Patient number55 | 2
  Patient number60 | 2.5
  Patient number64 | 2
  Patient number68 | 2
  Patient number69 | 2.5
  Patient number70 | 2
  Patient number73 | 2
  Patient number77 | 2
  Patient number78 | 2
  Patient number81 | 2.5

52. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Remifentanil After Intranasal Dexmedetomidine Before Inserting Operative Laryngoscope
Description: Predicted effect-site concentrations of remifentanil after intranasal dexmedetomidine before inserting operative laryngoscope.
  Remifentanil was infused to achieve a TCI plasma concentration of 3.0 ng∙ml-1 using the Minto pharmacokinetic model 24 and then adjusted to maintain the systolic blood pressure (SBP) at 25% of the pre-operative value and the HR at less than 90 bpm. To maintain a neuromuscular blockade, 0.15 mg∙kg-1 increments of rocuronium were infused upon observation of the first twitch in a train-of-four response with the nerve stimulator
Time Frame: 1 day
Measure: Number; unit: ng/ml
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
ng/ml
  Patient number2 | 2
  Patient number3 | 2
  Patient number5 | 2
  Patient number6 | 2
  Patient number7 | 2
  Patient number9 | 2
  Patient number10 | 2
  Patient number11 | 2
  Patient number18 | 2
  Patient number24 | 2
  Patient number25 | 2
  Patient number28 | 2
  Patient number29 | 2
  Patient number31 | 2
  Patient number33 | 2
  Patient number36 | 2
  Patient number38 | 2
  Patient number40 | 2
  Patient number44 | 2
  Patient number46 | 2
  Patient number50 | 2
  Patient number52 | 2
  Patient number53 | 2
  Patient number56 | 2
  Patient number57 | 2
  Patient number58 | 2
  Patient number59 | 2
  Patient number61 | 2
  Patient number62 | 2
  Patient number63 | 2
  Patient number65 | 2
  Patient number66 | 2
  Patient number67 | 2
  Patient number71 | 2
  Patient number72 | 2
  Patient number74 | 2
  Patient number75 | 2
  Patient number76 | 2
  Patient number79 | 2
  Patient number80 | 2

53. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Remifentanil After Intranasal Placebo on Removal of Operative Laryngoscope
Description: Predicted effect-site concentrations of remifentanil after intranasal placebo on removal of operative laryngoscope.
  Remifentanil was infused to achieve a TCI plasma concentration of 3.0 ng∙ml-1 using the Minto pharmacokinetic model 24 and then adjusted to maintain the systolic blood pressure (SBP) at 25% of the pre-operative value and the HR at less than 90 bpm. To maintain a neuromuscular blockade, 0.15 mg∙kg-1 increments of rocuronium were infused upon observation of the first twitch in a train-of-four response with the nerve stimulator
Time Frame: 1 day
Measure: Number; unit: ng/ml
Arm/Group | Placebo
Number analyzed (Participants) | 41
ng/ml
  Patient number1 | 2.5
  Patient number4 | 3
  Patient number8 | 4
  Patient number12 | 5
  Patient number13 | 4
  Patient number14 | 5
  Patient number15 | 2
  Patient number16 | 4
  Patient number17 | 2
  Patient number19 | 2
  Patient number20 | 2.5
  Patient number21 | 2
  Patient number22 | 2.5
  Patient number23 | 2.5
  Patient number26 | 4.5
  Patient number27 | 4.5
  Patient number30 | 2
  Patient number32 | 4
  Patient number34 | 2
  Patient number35 | 2.5
  Patient number37 | 2.5
  Patient number39 | 4.5
  Patient number41 | 5
  Patient number42 | 3
  Patient number43 | 2
  Patient number45 | 3.5
  Patient number47 | 5
  Patient number48 | 2
  Patient number49 | 3
  Patient number51 | 3.5
  Patient number54 | 2.5
  Patient number55 | 2
  Patient number60 | 3
  Patient number64 | 2.5
  Patient number68 | 2
  Patient number69 | 2
  Patient number70 | 2.5
  Patient number73 | 4
  Patient number77 | 2
  Patient number78 | 2
  Patient number81 | 3

54. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Remifentanil After Intranasal Dexmedetomidine on Removal of Operative Laryngoscope
Description: Predicted effect-site concentrations of remifentanil after intranasal dexmedetomidine on removal of operative laryngoscope.
  Remifentanil was infused to achieve a TCI plasma concentration of 3.0 ng∙ml-1 using the Minto pharmacokinetic model 24 and then adjusted to maintain the systolic blood pressure (SBP) at 25% of the pre-operative value and the HR at less than 90 bpm. To maintain a neuromuscular blockade, 0.15 mg∙kg-1 increments of rocuronium were infused upon observation of the first twitch in a train-of-four response with the nerve stimulator
Time Frame: 1 day
Measure: Number; unit: ng/ml
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
ng/ml
  Patient number2 | 2
  Patient number3 | 2
  Patient number5 | 2
  Patient number6 | 2
  Patient number7 | 2.5
  Patient number9 | 2.5
  Patient number10 | 2.5
  Patient number11 | 2
  Patient number18 | 3
  Patient number24 | 2.5
  Patient number25 | 2
  Patient number28 | 2
  Patient number29 | 3
  Patient number31 | 3
  Patient number33 | 2
  Patient number36 | 2
  Patient number38 | 2
  Patient number40 | 2
  Patient number44 | 3
  Patient number46 | 2.5
  Patient number50 | 3
  Patient number52 | 2
  Patient number53 | 2
  Patient number56 | 2
  Patient number57 | 2.5
  Patient number58 | 4
  Patient number59 | 2
  Patient number61 | 4
  Patient number62 | 2
  Patient number63 | 2
  Patient number65 | 2
  Patient number66 | 2
  Patient number67 | 3
  Patient number71 | 2
  Patient number72 | 3.5
  Patient number74 | 3
  Patient number75 | 3
  Patient number76 | 2
  Patient number79 | 2
  Patient number80 | 2

55. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Remifentanil After Intranasal Placebo at Return of Spontaneous Breathing
Description: Predicted effect-site concentrations of remifentanil after intranasal placebo at return of spontaneous breathing.
  Remifentanil was infused to achieve a TCI plasma concentration of 3.0 ng∙ml-1 using the Minto pharmacokinetic model 24 and then adjusted to maintain the systolic blood pressure (SBP) at 25% of the pre-operative value and the HR at less than 90 bpm. To maintain a neuromuscular blockade, 0.15 mg∙kg-1 increments of rocuronium were infused upon observation of the first twitch in a train-of-four response with the nerve stimulator
Time Frame: 1 day
Measure: Number; unit: ng/ml
Arm/Group | Placebo
Number analyzed (Participants) | 41
ng/ml
  Patient number1 | 0.98
  Patient number4 | 1.03
  Patient number8 | 1
  Patient number12 | 1.3
  Patient number13 | 0.8
  Patient number14 | 1.3
  Patient number15 | 0.27
  Patient number16 | 0.7
  Patient number17 | 0.35
  Patient number19 | 0.3
  Patient number20 | 0.98
  Patient number21 | 0.35
  Patient number22 | 0.54
  Patient number23 | 0.6
  Patient number26 | 0.8
  Patient number27 | 0.7
  Patient number30 | 0.2
  Patient number32 | 0.9
  Patient number34 | 0.5
  Patient number35 | 0.6
  Patient number37 | 0.6
  Patient number39 | 1
  Patient number41 | 1.1
  Patient number42 | 0.6
  Patient number43 | 0.5
  Patient number45 | 1.1
  Patient number47 | 1.3
  Patient number48 | 0.6
  Patient number49 | 1.28
  Patient number51 | 0.78
  Patient number54 | 1.4
  Patient number55 | 0.16
  Patient number60 | 1
  Patient number64 | 0.41
  Patient number68 | 0.5
  Patient number69 | 0.6
  Patient number70 | 1.2
  Patient number73 | 0.9
  Patient number77 | 0.4
  Patient number78 | 0.5
  Patient number81 | 0.8

56. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Remifentanil After Intranasal Dexmedetomidine at Return of Spontaneous Breathing
Description: Predicted effect-site concentrations of remifentanil after intranasal dexmedetomidine at return of spontaneous breathing.
  Remifentanil was infused to achieve a TCI plasma concentration of 3.0 ng∙ml-1 using the Minto pharmacokinetic model 24 and then adjusted to maintain the systolic blood pressure (SBP) at 25% of the pre-operative value and the HR at less than 90 bpm. To maintain a neuromuscular blockade, 0.15 mg∙kg-1 increments of rocuronium were infused upon observation of the first twitch in a train-of-four response with the nerve stimulator
Time Frame: 1 day
Measure: Number; unit: ng/ml
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
ng/ml
  Patient number2 | 0.6
  Patient number3 | 0.7
  Patient number5 | 0.56
  Patient number6 | 0.6
  Patient number7 | 0.6
  Patient number9 | 0.6
  Patient number10 | 0.83
  Patient number11 | 0.4
  Patient number18 | 0.75
  Patient number24 | 0.18
  Patient number25 | 0.3
  Patient number28 | 0.7
  Patient number29 | 0.6
  Patient number31 | 0.47
  Patient number33 | 0.35
  Patient number36 | 0.6
  Patient number38 | 0.4
  Patient number40 | 0.4
  Patient number44 | 0.47
  Patient number46 | 0.71
  Patient number50 | 0.75
  Patient number52 | 0.5
  Patient number52 | 0.7
  Patient number56 | 0.5
  Patient number57 | 0.56
  Patient number58 | 1.28
  Patient number59 | 0.35
  Patient number61 | 1.28
  Patient number62 | 0.5
  Patient number63 | 0.2
  Patient number65 | 0.3
  Patient number66 | 0.5
  Patient number67 | 0.41
  Patient number71 | 0.6
  Patient number72 | 0.78
  Patient number74 | 0.6
  Patient number75 | 1
  Patient number76 | 0.27
  Patient number79 | 0.5
  Patient number80 | 0.09

57. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Remifentanil After Intranasal Placebo at Emergence
Description: Predicted effect-site concentrations of remifentanil after intranasal placebo at emergence.
  Remifentanil was infused to achieve a TCI plasma concentration of 3.0 ng∙ml-1 using the Minto pharmacokinetic model 24 and then adjusted to maintain the systolic blood pressure (SBP) at 25% of the pre-operative value and the HR at less than 90 bpm. To maintain a neuromuscular blockade, 0.15 mg∙kg-1 increments of rocuronium were infused upon observation of the first twitch in a train-of-four response with the nerve stimulator
Time Frame: 1 day
Measure: Number; unit: ng/ml
Arm/Group | Placebo
Number analyzed (Participants) | 41
ng/ml
  Patient number1 | 0.54
  Patient number4 | 0.47
  Patient number8 | 0.8
  Patient number12 | 1.1
  Patient number13 | 0.4
  Patient number14 | 0.7
  Patient number15 | 0.04
  Patient number16 | 0.3
  Patient number17 | 0.13
  Patient number19 | 0.1
  Patient number20 | 0.14
  Patient number21 | 0.16
  Patient number22 | 0.37
  Patient number23 | 0.41
  Patient number26 | 0.4
  Patient number27 | 0.3
  Patient number30 | 0.16
  Patient number32 | 0.4
  Patient number34 | 0.14
  Patient number35 | 0.29
  Patient number37 | 0.37
  Patient number39 | 0.4
  Patient number41 | 0.4
  Patient number42 | 0.28
  Patient number43 | 0.16
  Patient number45 | 0.3
  Patient number47 | 0.8
  Patient number48 | 0.4
  Patient number49 | 0.28
  Patient number51 | 0.2
  Patient number54 | 0.98
  Patient number55 | 0.04
  Patient number60 | 0.32
  Patient number64 | 0.29
  Patient number68 | 0.27
  Patient number69 | 0.24
  Patient number70 | 0.29
  Patient number73 | 0.1
  Patient number77 | 0.2
  Patient number78 | 0.02
  Patient number81 | 0.34

58. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Remifentanil After Intranasal Dexmedetomidine at Emergence
Description: Predicted effect-site concentrations of remifentanil after intranasal dexmedetomidine at emergence.
  Remifentanil was infused to achieve a TCI plasma concentration of 3.0 ng∙ml-1 using the Minto pharmacokinetic model 24 and then adjusted to maintain the systolic blood pressure (SBP) at 25% of the pre-operative value and the HR at less than 90 bpm. To maintain a neuromuscular blockade, 0.15 mg∙kg-1 increments of rocuronium were infused upon observation of the first twitch in a train-of-four response with the nerve stimulator
Time Frame: 1 day
Measure: Number; unit: ng/ml
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
ng/ml
  Patient number2 | 0.27
  Patient number3 | 0.18
  Patient number5 | 0.2
  Patient number6 | 0.27
  Patient number7 | 0.18
  Patient number9 | 0.32
  Patient number10 | 0.23
  Patient number11 | 0.27
  Patient number18 | 0.37
  Patient number24 | 0.1
  Patient number25 | 0.18
  Patient number28 | 0.24
  Patient number29 | 0.04
  Patient number31 | 0.23
  Patient number33 | 0.1
  Patient number36 | 0.24
  Patient number38 | 0.11
  Patient number40 | 0.14
  Patient number44 | 0.02
  Patient number46 | 0.29
  Patient number50 | 0.28
  Patient number52 | 0.3
  Patient number53 | 0.3
  Patient number56 | 0.1
  Patient number57 | 0.2
  Patient number58 | 0.3
  Patient number59 | 0.14
  Patient number61 | 0.2
  Patient number62 | 0.1
  Patient number63 | 0.06
  Patient number65 | 0.1
  Patient number66 | 0.24
  Patient number67 | 0.18
  Patient number71 | 0.3
  Patient number72 | 0.4
  Patient number74 | 0.47
  Patient number75 | 0.28
  Patient number76 | 0.2
  Patient number79 | 0.18
  Patient number80 | 0.05

59. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Remifentanil After Intranasal Placebo at Extubation
Description: Predicted effect-site concentrations of remifentanil after intranasal placebo at extubation.
  Remifentanil was infused to achieve a TCI plasma concentration of 3.0 ng∙ml-1 using the Minto pharmacokinetic model 24 and then adjusted to maintain the systolic blood pressure (SBP) at 25% of the pre-operative value and the HR at less than 90 bpm. To maintain a neuromuscular blockade, 0.15 mg∙kg-1 increments of rocuronium were infused upon observation of the first twitch in a train-of-four response with the nerve stimulator
Time Frame: 1 day
Measure: Number; unit: ng/ml
Arm/Group | Placebo
Number analyzed (Participants) | 41
ng/ml
  Patient number1 | 0.41
  Patient number4 | 0.37
  Patient number8 | 0.7
  Patient number12 | 0.8
  Patient number13 | 0.3
  Patient number14 | 0.5
  Patient number15 | 0.03
  Patient number16 | 0.2
  Patient number17 | 0.1
  Patient number19 | 0.08
  Patient number20 | 0.11
  Patient number21 | 0.13
  Patient number22 | 0.29
  Patient number23 | 0.37
  Patient number26 | 0.3
  Patient number27 | 0.22
  Patient number30 | 0.11
  Patient number32 | 0.3
  Patient number34 | 0.1
  Patient number35 | 0.18
  Patient number37 | 0.29
  Patient number39 | 0.3
  Patient number41 | 0.3
  Patient number42 | 0.23
  Patient number43 | 0.14
  Patient number45 | 0.2
  Patient number47 | 0.7
  Patient number48 | 0.35
  Patient number49 | 0.23
  Patient number51 | 0.1
  Patient number54 | 0.6
  Patient number55 | 0.04
  Patient number60 | 0.26
  Patient number64 | 0.26
  Patient number68 | 0.2
  Patient number69 | 0.14
  Patient number70 | 0.23
  Patient number73 | 0.1
  Patient number77 | 0.16
  Patient number78 | 0.02
  Patient number81 | 0.26

60. Other Pre Specified Outcome: Predicted Effect-site Concentrations of Remifentanil After Intranasal Dexmedetomidine at Extubation
Description: Predicted effect-site concentrations of remifentanil after intranasal dexmedetomidine at extubation.
  Remifentanil was infused to achieve a TCI plasma concentration of 3.0 ng∙ml-1 using the Minto pharmacokinetic model 24 and then adjusted to maintain the systolic blood pressure (SBP) at 25% of the pre-operative value and the HR at less than 90 bpm. To maintain a neuromuscular blockade, 0.15 mg∙kg-1 increments of rocuronium were infused upon observation of the first twitch in a train-of-four response with the nerve stimulator
Time Frame: 1 day
Measure: Number; unit: ng/ml
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
ng/ml
  Patient number2 | 0.24
  Patient number3 | 0.16
  Patient number5 | 0.16
  Patient number6 | 0.2
  Patient number7 | 0.14
  Patient number9 | 0.29
  Patient number14 | 0.23
  Patient number11 | 0.2
  Patient number18 | 0.28
  Patient number24 | 0.08
  Patient number25 | 0.14
  Patient number28 | 0.18
  Patient number29 | 0.03
  Patient number31 | 0.18
  Patient number33 | 0.07
  Patient number36 | 0.13
  Patient number38 | 0.08
  Patient number40 | 0.11
  Patient number44 | 0.01
  Patient number46 | 0.23
  Patient number50 | 0.23
  Patient number52 | 0.27
  Patient number53 | 0.27
  Patient number56 | 0.08
  Patient number57 | 0.17
  Patient number58 | 0.2
  Patient number59 | 0.1
  Patient number61 | 0.1
  Patient number62 | 0.07
  Patient number63 | 0.04
  Patient number65 | 0.06
  Patient number66 | 0.18
  Patient number67 | 0.11
  Patient number71 | 0.27
  Patient number72 | 0.4
  Patient number74 | 0.41
  Patient number75 | 0.26
  Patient number76 | 0.16
  Patient number79 | 0.14
  Patient number80 | 0.04

61. Other Pre Specified Outcome: HR in the Placebo Group Before Intranasal Drugs
Description: HR in the placebo group Before Intranasal Drugs HR was monitored by fiber-optic pulse oximetry during patient transfer from the ward to the operating room
Time Frame: 1 day
Measure: Number; unit: bpm
Arm/Group | Placebo
Number analyzed (Participants) | 41
bpm
  Patient number1 | 65
  Patient number4 | 77
  Patient number8 | 61
  Patient number12 | 80
  Patient number13 | 67
  Patient number14 | 75
  Patient number15 | 55
  Patient number16 | 65
  Patient number17 | 78
  Patient number19 | 57
  Patient number20 | 76
  Patient number21 | 85
  Patient number22 | 69
  Patient number23 | 71
  Patient number26 | 75
  Patient number27 | 65
  Patient number30 | 100
  Patient number32 | 83
  Patient number34 | 55
  Patient number35 | 72
  Patient number37 | 75
  Patient number39 | 75
  Patient number41 | 120
  Patient number42 | 59
  Patient number43 | 89
  Patient number45 | 90
  Patient number47 | 74
  Patient number48 | 63
  Patient number49 | 88
  Patient number51 | 56
  Patient number54 | 75
  Patient number55 | 63
  Patient number60 | 82
  Patient number64 | 80
  Patient number68 | 65
  Patient number69 | 63
  Patient number70 | 64
  Patient number73 | 65
  Patient number77 | 63
  Patient number78 | 55
  Patient number81 | 72

62. Other Pre Specified Outcome: HR in the Dexmedetomidine Group Before Intranasal Drugs
Description: HR in the dexmedetomidine group Before Intranasal Drugs . HR was monitored by fiber-optic pulse oximetry during patient transfer from the ward to the operating room
Time Frame: 1 day
Measure: Number; unit: bpm
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
bpm
  Patient number2 | 73
  Patient number3 | 68
  Patient number5 | 80
  Patient number6 | 80
  Patient number7 | 67
  Patient number9 | 70
  Patient number10 | 69
  Patient number11 | 70
  Patient number18 | 75
  Patient number24 | 80
  Patient number25 | 75
  Patient number28 | 87
  Patient number29 | 73
  Patient number33 | 60
  Patient number33 | 90
  Patient number36 | 73
  Patient number38 | 58
  Patient number40 | 66
  Patient number44 | 80
  Patient number46 | 85
  Patient number50 | 71
  Patient number52 | 79
  Patient number53 | 69
  Patient number56 | 75
  Patient number57 | 76
  Patient number58 | 61
  Patient number59 | 70
  Patient number61 | 55
  Patient number62 | 97
  Patient number63 | 68
  Patient number65 | 65
  Patient number66 | 65
  Patient number67 | 67
  Patient number71 | 80
  Patient number72 | 55
  Patient number74 | 62
  Patient number75 | 69
  Patient number76 | 80
  Patient number79 | 55
  Patient number80 | 69

63. Other Pre Specified Outcome: HR in the Placebo Group at Pre-induction
Description: HR in the placebo group at pre-induction. HR was monitored by fiber-optic pulse oximetry during patient transfer from the ward to the operating room
Time Frame: 1 day
Measure: Number; unit: bpm
Arm/Group | Placebo
Number analyzed (Participants) | 41
bpm
  Patient number1 | 76
  Patient number4 | 85
  Patient number8 | 63
  Patient number12 | 80
  Patient number13 | 53
  Patient number14 | 79
  Patient number15 | 62
  Patient number16 | 72
  Patient number17 | 70
  Patient number19 | 59
  Patient number20 | 74
  Patient number21 | 73
  Patient number22 | 90
  Patient number23 | 82
  Patient number26 | 78
  Patient number27 | 61
  Patient number30 | 92
  Patient number32 | 85
  Patient number34 | 54
  Patient number35 | 66
  Patient number37 | 75
  Patient number39 | 60
  Patient number41 | 94
  Patient number42 | 72
  Patient number43 | 85
  Patient number45 | 87
  Patient number47 | 81
  Patient number48 | 61
  Patient number49 | 72
  Patient number51 | 53
  Patient number54 | 70
  Patient number55 | 72
  Patient number60 | 78
  Patient number64 | 75
  Patient number68 | 70
  Patient number69 | 69
  Patient number70 | 62
  Patient number73 | 69
  Patient number77 | 66
  Patient number78 | 55
  Patient number81 | 72

64. Other Pre Specified Outcome: HR in the Dexmedetomidine Group at Pre-induction
Description: HR in the dexmedetomidine group at pre-induction. HR was monitored by fiber-optic pulse oximetry during patient transfer from the ward to the operating room
Time Frame: 1 day
Measure: Number; unit: bpm
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
bpm
  Patient number2 | 62
  Patient number3 | 62
  Patient number5 | 93
  Patient number6 | 70
  Patient number7 | 53
  Patient number9 | 75
  Patient number10 | 62
  Patient number11 | 55
  Patient number18 | 59
  Patient number24 | 68
  Patient number25 | 60
  Patient number28 | 88
  Patient number29 | 66
  Patient number31 | 64
  Patient number33 | 69
  Patient number36 | 61
  Patient number38 | 48
  Patient number40 | 55
  Patient number44 | 76
  Patient number46 | 80
  Patient number50 | 70
  Patient number52 | 72
  Patient number53 | 64
  Patient number56 | 68
  Patient number57 | 63
  Patient number58 | 54
  Patient number59 | 54
  Patient number61 | 63
  Patient number62 | 83
  Patient number63 | 73
  Patient number65 | 68
  Patient number66 | 66
  Patient number67 | 61
  Patient number71 | 53
  Patient number72 | 64
  Patient number74 | 55
  Patient number75 | 67
  Patient number76 | 71
  Patient number79 | 62
  Patient number80 | 65

65. Other Pre Specified Outcome: Number of Participants With VAS >50
Description: Patients with postoperative analgesia in two groups. analgesic requests within 2 h after extubation were recorded. An investigator who was blinded from the grouping asked the patients to mark their pain level on a 0-100 visual analogue scale (VAS). A VAS higher than 50 was considered a worse outcome and need to be treated with intravenous 40 mg of parecoxib.
Time Frame: 1 day
Measure: Number; unit: Number of Participants with VAS >50
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 40 | 41
Number of Participants with VAS >50 | 5 | 15

66. Other Pre Specified Outcome: Patients With Postoperative Nausea in Two Groups
Description: Patients With postoperative nausea in Two Groups. Nausea or vomiting was treated with 4 mg of intravenous ondansetron.
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 40 | 41
participants | 1 | 3

67. Other Pre Specified Outcome: Patients With Postoperative Vomiting in Two Groups
Description: Patients With postoperative vomiting in Two Groups. Nausea or vomiting was treated with 4 mg of intravenous ondansetron.
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 40 | 41
participants | 0 | 1

68. Other Pre Specified Outcome: Patients With Postoperative Shivering in Two Groups
Description: Patients With postoperative shivering in Two Groups. the occurrence of postoperative shivering
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 40 | 41
participants | 1 | 4

69. Other Pre Specified Outcome: Patients With Intra-operative Awareness in Two Groups
Description: Patients With intra-operative awareness in Two Groups. patients receiving intranasal placebo or dexmedetomidine
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 40 | 41
participants | 0 | 0

70. Other Pre Specified Outcome: Visual Analogue Scale (VAS) in the Placebo Group
Description: An investigator who was blinded from the grouping asked the patients to mark their pain level on a 0-100 visual analogue scale (VAS). A VAS higher than 50 was considered a worse outcome and need to be treated with intravenous 40 mg of parecoxib.
Time Frame: 1 day
Measure: Number; unit: units on a scale
Arm/Group | Placebo
Number analyzed (Participants) | 41
units on a scale
  Patient number1 | 80
  Patient number4 | 20
  Patient number8 | 20
  Patient number12 | 80
  Patient number13 | 80
  Patient number14 | 80
  Patient number15 | 20
  Patient number16 | 0
  Patient number17 | 80
  Patient number19 | 20
  Patient number20 | 80
  Patient number21 | 20
  Patient number22 | 20
  Patient number23 | 20
  Patient number26 | 20
  Patient number27 | 20
  Patient number30 | 80
  Patient number32 | 20
  Patient number34 | 20
  Patient number35 | 20
  Patient number37 | 20
  Patient number39 | 20
  Patient number41 | 20
  Patient number42 | 20
  Patient number43 | 0
  Patient number45 | 20
  Patient number47 | 80
  Patient number48 | 80
  Patient number49 | 80
  Patient number51 | 20
  Patient number54 | 20
  Patient number55 | 80
  Patient number60 | 80
  Patient number64 | 80
  Patient number68 | 20
  Patient number69 | 80
  Patient number70 | 20
  Patient number73 | 80
  Patient number77 | 0
  Patient number78 | 20
  Patient number81 | 20

71. Other Pre Specified Outcome: Visual Analogue Scale (VAS) in the Dexmedetomidine (DEX) Group
Description: as for outcome 70
Time Frame: 1 day
Measure: Number; unit: units on a scale
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 40
units on a scale
  Patient number2 | 20
  Patient number3 | 20
  Patient number5 | 20
  Patient number6 | 20
  Patient number7 | 80
  Patient number9 | 20
  Patient number10 | 20
  Patient number11 | 20
  Patient number18 | 20
  Patient number24 | 20
  Patient number25 | 20
  Patient number28 | 20
  Patient number29 | 20
  Patient number31 | 20
  Patient number33 | 0
  Patient number36 | 20
  Patient number38 | 0
  Patient number40 | 80
  Patient number44 | 80
  Patient number46 | 20
  Patient number50 | 20
  Patient number52 | 20
  Patient number53 | 20
  Patient number56 | 20
  Patient number57 | 20
  Patient number58 | 20
  Patient number59 | 20
  Patient number61 | 20
  Patient number62 | 20
  Patient number63 | 20
  Patient number65 | 20
  Patient number66 | 20
  Patient number67 | 20
  Patient number71 | 80
  Patient number72 | 20
  Patient number74 | 20
  Patient number75 | 0
  Patient number76 | 20
  Patient number79 | 20
  Patient number80 | 20

72. Secondary Outcome: Anxiety Score of Patients Receiving Intranasal Placebo or Dexmedetomidine
Description: 4-point anxiety score:
  1. = combative
  2. = anxious
  3. = calm
  4. = amiable. Anxiety score >2 was considered to be better for the preoperative patients.
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 40 | 41
units on a scale
  Before intranasal drugs | 3 [2 to 3] | 3 [2 to 3]
  Pre-induction | 3 [3 to 4] | 3 [2 to 3]

73. Secondary Outcome: Systolic Blood Pressure（SBP）of Patients Receiving Intranasal Placebo or Dexmedetomidine
Description: Systolic blood pressure（SBP）of Patients Receiving Intranasal Placebo or Dexmedetomidine.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 40 | 41
mmHg
  Before intranasal drops | 120.8684 (2.07579) | 116.8462 (1.71622)
  On arrival at operating room | 120.5641 (2.96079) | 126.875 (2.6373)
  At pre-induction | 117.725 (2.73322) | 122.6 (2.5285)
  After tracheal intubation | 121.57 (13.97) | 119.52 (14.94)
  After inserting operative laryngoscope | 130.00 (21.24) | 123.65 (19.60)
  After removal of laryngoscope | 126.33 (15.96) | 123.39 (10.16)
  On arrival at PACU | 128.52 (17.81) | 123.90 (14.61)
  At emergency | 132.76 (18.20) | 130.71 (16.67)
  After tracheal extubation | 136.76 (21.11) | 132.13 (19.14)
  Before leaving PACU | 130.00 (14.81) | 127.97 (13.41)

74. Secondary Outcome: Number of Participants With Satisfaction Score <2
Description: Patient satisfaction scores using a 3-point satisfaction score (1 = highly satisfactory, 2 = acceptable, and 3 = unacceptable) were collected when patients were discharged from the post-anesthesia care unit (PACU).
  Satisfaction score <2 was considered to be better for the patient
Time Frame: 1 day
Measure: Number; unit: participant
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 40 | 41
participant | 34 | 25

75. Secondary Outcome: Perioperative Bradycardia Episodes
Description: Bradycardia was defined as heart rate (HR) <45 bpm for more than 10 s.
Time Frame: 1 day
Measure: Number; unit: participant
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 40 | 41
participant
  Bradycardiac episode:Pre-induction | 2 | 0
  Bradycardiac episode:After intubation | 1 | 1
  Bradycardiac episode:Intra-operative | 3 | 5
  Bradycardiac episode:After extubation | 7 | 5

76. Secondary Outcome: Perioperative Tachycardia Episodes
Description: Tachycardia was defined as heart rate (HR) >100 bpm for more than 10 s.
Time Frame: 1 day
Measure: Number; unit: participant
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 40 | 41
participant
  Tachycardiac episode:Pre-induction | 0 | 0
  Tachycardiac episode:After intubation | 1 | 8
  Tachycardiac episode:Intra-operative | 5 | 11
  Tachycardiac episode:After extubation | 2 | 9

77. Secondary Outcome: Perioperative Hypotension Episodes
Description: Hypotension was defined as systolic blood pressure (SBP) decreased more than 30% of the pre-operative value for more than 1 min.
Time Frame: 1 day
Measure: Number; unit: participant
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 40 | 41
participant
  Hypotensive episode:Pre-induction | 0 | 2
  Hypotensive episode:After intubation | 3 | 4
  Hypotensive episode:Post-induction | 3 | 4
  Hypotensive episode:After extubation | 1 | 0

78. Secondary Outcome: Perioperative Hypertonsion Episodes
Description: Hypertension was defined as systolic blood pressure (SBP) increased 130% of the pre-operative value for more than 1 min.
Time Frame: 1 day
Measure: Number; unit: participant
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 40 | 41
participant
  Hypertensive episode:Pre-induction | 1 | 0
  Hypertensive episode:After intubation | 6 | 0
  Hypertensive episode:Intra-operative | 6 | 5
  Hypertensive episode:After extubation | 14 | 5

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Dexmedetomidine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 20/40 | 34/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine (N=40) | Placebo (N=41)
Number of patients with persisted hypotension (Cardiac disorders) | 0 (0) | 0 (0) — Number of patients with persisted hypotension after administration of ephedrine more than 30 mg.
Number of patients with persisted bradycardia (Cardiac disorders) | 0 (0) | 0 (0) — Number of patients with persisted bradycardia after administration of atropine more than 2.0 mg.
intraoperative awareness (Nervous system disorders) | 0 (0) | 0 (0) — On the first post-operative day, follow-up interviews to determine intra-operative recall of the patients.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine (N=40) | Placebo (N=41)
Episodes of hypertension (Cardiac disorders) | 9 (9) | 16 (16) — Systolic blood pressure (SBP) increased 130% of the pre-operative value for more than 1 min.
Episodes of hypotension (Cardiac disorders) | 1 (1) | 0 (0) — Systolic blood pressure (SBP) decreased more than 30% of the pre-operative value for more than 1 min.
Episodes of tachycardia (Cardiac disorders) | 7 (7) | 20 (20) — Heart rate (HR) >100 bpm for more than 10 s.
Episodes of bradycardia (Cardiac disorders) | 8 (8) | 10 (10) — Heart rate (HR) <45 bpm for more than 10 s.
Episodes of Respiratory depression (Reproductive system and breast disorders) | 5 (5) | 11 (11) — Respiratory rate (RR) <8 bpm and oxygen saturation (SpO2) <90%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No